

# Protocol Cover Page

Protocol Title: An Extension Protocol for Virologically Suppressed Subjects Who Successfully

Completed PRO140\_CD03 Study

Protocol Number: PRO 140\_CD03 Extension

Version: 5.0

**Document Date: 30-Mar-2021** 

NCT Number: NCT05271370



# An Extension Protocol for Virologically Suppressed Subjects Who Successfully Completed PRO140\_CD03 Study

Protocol Number: PRO 140\_CD03 Extension

Version: 5.0

Date: 30-Mar-2021

Sponsor: CytoDyn, Inc.

1111 Main Street, Suite 660 Vancouver, Washington 98660 (360) 980-8524-Work (360) 980-8549-Fax

www.cytodyn.com

# **Confidentiality Statement**

This document is a confidential communication of CytoDyn, Inc. It is provided for the conduct of a clinical research study. The information contained in this document is confidential and, except to the extent necessary to obtain informed consent or IEC/IRB approval, cannot be disclosed unless required by governmental regulation. Persons to whom any portion of the contents of this document is disclosed must be informed that the information is confidential and may not be further disclosed by them.




# PROTOCOL APPROVAL PAGE

Protocol Number: PRO 140\_CD03 Extension

Version: 5.0

Date: 30-Mar-2021

### PROTOCOL APPROVAL FOR USE

I have read the protocol and the appendices and agree that it contains all relevant information required to meet FDA, GCP and all applicable regulatory guidelines and statutes.

| Prepared by: | |
|--------------|------|
| | Date |
| Reviewed by: | |
| | Date |
| | Date |
| | Date |
| Approved by: | Date |




# **INVESTIGATOR'S SIGNATURE PAGE**

Protocol Number: PRO 140\_CD03 Extension

Version: 5.0

Date: 30-Mar-2021

### **INVESTIGATOR'S SIGNATURE**

I have read the protocol specified above and agree to participate in and comply with the procedures, as outlined herein for the conduct of this clinical trial. I also agree to comply with the applicable US Food and Drug Administration (FDA) regulations and Investigational Review Board (IRB) requirements for testing on human subjects. I agree to ensure that the requirements for obtaining informed consent are met.

| Principal Investigator's Signature | Date |
|------------------------------------|------|
| Print Name | |
| Address | |
| ridicos | |
| Site Number | |




# **SPONSOR INFORMATION**

CytoDyn, Inc.

1111 Main Street, Suite 660 Vancouver, Washington 98660 (360) 980-8524-Work (360) 980-8549-Fax www.cytodyn.com

# **CONTRACT RESEARCH ORGANIZATION INFORMATION**






PROTOCOL SYNOPSIS

| Name of Sponsor:<br>CytoDyn, Inc. | |
|---|---|
| Name of Study Product: PRO 140 (Humanized monoclonal antibody to CCR5) | |
| Protocol Number: | Indication: |
| PRO 140 _CD03 Extension | Human Immunodeficiency Virus Type-1 (HIV-1) Infection |

# Title of Study:

An Extension Protocol for Virologically Suppressed Subjects who Successfully Completed PRO140\_CD03 Study

Study Center(s): Site(s) participating in the PRO140\_CD03 Protocol

| Planned Number of Subjects: | Study Development Phase: |
|-----------------------------|--------------------------|
| Up to 300 subjects | Phase-2b/3 |

### **Study Population:**

Study population includes treatment-experienced HIV-infected patients with CCR5-tropic virus who successfully complete 48 weeks of treatment with PRO140 350mg, 525mg, or 700mg SC monotherapy under CD03 study.

**Objective:** The objective is to assess the long-term safety of using PRO 140 350mg, 525mg, or 700mg SC as single-agent maintenance therapy for the chronic suppression of CCR5-tropic HIV-1 infection.

### **Outcome Measures:**

### **Primary Outcome Measures:**

- Assess the long term clinical safety of PRO 140 350mg, 525, or 700 mg monotherapy regimen
- Proportion of participants experiencing virologic failure for all subjects and within each treatment group

# **Secondary Outcome Measures:**

- Time to virologic failure for all subjects and within each treatment group
- Proportion of participants achieving viral re-suppression (HIV-1 RNA < 50 copies/mL) after experiencing virologic failure for all subjects and within each treatment group
- Time to achieving viral re-suppression (HIV-1 RNA < 50 copies/mL) after experiencing virologic failure for all subjects and within each treatment group
- Proportion of virologic failure subjects achieving viral re-suppression with re-initiation of previous baseline antiretroviral regimen for all subjects and within each treatment group
- Mean change in CD4 cell count, at each visit within the Treatment Phase for all subjects and within
  each treatment group

### Safety Assessments:






| Name | of | Sn | On | co |
|-------|----|----|-----|-----|
| Maine | OI | op | UII | 190 |

CytoDyn, Inc.

### Name of Study Product:

PRO 140 (Humanized monoclonal antibody to CCR5)

**Protocol Number:** 

Indication:

PRO 140 CD03 Extension

Human Immunodeficiency Virus Type-1 (HIV-1) Infection

- Tolerability of repeated subcutaneous administration of PRO 140 350mg, 525mg, or 700mg as assessed by investigator-evaluation of injection site reactions for all subjects and within each treatment group
- Frequency of Grade 2, 3 or 4 adverse events as defined by the DAIDS Adverse Event scale
- Frequency of Treatment-emergent serious adverse events

### Trial Design:

This study is a Phase 2b/3 multi-center extension study designed to evaluate the long term antiviral activity, safety, and tolerability of the strategy of continuing PRO 140 350mg, 525mg, or 700mg SC monotherapy to maintain viral suppression after initial 48 weeks in virologically suppressed subjects.

Consenting subjects will continue weekly PRO 140 350mg, 525mg, or 700mg monotherapy during the Treatment Extension Phase with the one week overlap of existing retroviral regimen and PRO 140 350mg, 525mg, or 700 mg at the end of the treatment in subjects who do not experience virologic failure.

The study will have three phases: Screening Phase, Treatment Extension Phase, and Follow-up Phase.

### Screening Phase (up to 21 days):

This phase is designed to determine whether subjects are eligible to proceed to the Treatment Extension Phase of the study. This phase consists of a series of screening assessments designed to determine eligibility. A written informed consent from the subject will be obtained by the Investigator or suitably qualified individual before the performance of any protocol-specific procedure.

Screening Phase will consist of screening visit that corresponds to Treatment Visit 46/47/48 under the PRO 140 CD 03 study, and potential subjects will continue receiving PRO 140 350mg, 525mg, or 700mg monotherapy during the Screening Phase.

Note: Subjects who intend and consent to participate in Treatment Extension study will not initiate ART Regimen therapy at T47.

# Treatment Extension Phase (weekly ±3 days):

Treatment Extension Phase begins with an evaluation of most recent results of laboratory samples collected during the Screening Phase (viral load and CD4 count). Subjects who meet all eligibility criteria, as per data gathered from Screening Phase will receive PRO 140 350mg, 525mg, or 700mg at first Treatment Extension Visit (TE1). All subjects who fail to meet eligibility criteria will be considered screen failures and exit the study without further evaluation.

The first Treatment Extension Visit (TE1) will take place within 10 days of last treatment visit under CD03 study (i.e. T48 visit), with weekly visits (± 3 days) thereafter.

CONFIDENTIAL. 



| Name of Sponsor:<br>CytoDyn, Inc. | |
|---|---|
| Name of Study Product:<br>PRO 140 (Humanized monoclonal antibo | dy to CCR5) |
| Protocol Number: PRO 140 CD03 Extension | Indication: Human Immunodeficiency Virus Type-1 (HIV-1) Infection |

Subjects will continue PRO 140 350mg, 525mg, 700mg monotherapy injections, administered by a qualified medical professional (MD, DO, PA, LPN, LVN, NP, RN, or CMA if state law permits) at clinic site or home visit or self-administered by subjects throughout the Treatment Extension Phase.

Subjects who receive PRO 140 350mg and experience virologic failure during the Treatment Extension Phase have the option of receiving PRO 140 525mg for the remainder of the Treatment Extension Phase or may reinitiate prior ART regimen (or an alternative regimen selected by their treating physician) at the discretion of the Investigator.

Subjects who receive PRO 140 525mg and experience virologic failure during the Treatment Extension Phase have the option of receiving PRO 140 700mg for remainder of the Treatment Extension Phase or may reinitiate prior ART regimen (or an alternative regimen selected by their treating physician at the discretion of the Investigator

Subjects receiving PRO 140 350 mg who do <u>not</u> elect to receive PRO 140 525mg, and subjects receiving PRO 140 525mg who do <u>not</u> elect to receive PRO 140 700mg of the Treatment Extension Phase, and all subjects receiving PRO 140 700 mg who experience virologic failure (defined as two consecutive HIV-1 RNA levels of  $\geq$  200 copies/mL) at any time during the Treatment Extension Phase, will undergo the Virologic Failure (VF) Visit assessments and then exit the Treatment Extension Phase to enter the Follow-up Phase of the study.

Subjects who do not experience virologic failure will complete the EOT assessments and then enter the Follow-up Phase of the study at the end of Treatment Extension Phase.

All study subjects will re-initiate their previous antiretroviral regimen or an alternative regimen selected by their treating physician:

- One week prior to the end of Treatment Extension Phase, or
- During the Treatment Extension Phase, if virologic failure occurs or have met any other criteria for discontinuation of study treatment as specified in Section 5.2.1 of the protocol.

Efficacy assessments will include viral load measurement and CD4 cell counts once every four weeks during the Treatment Extension Phase. Safety assessments will consist of determining and recording all AEs and SAEs; laboratory evaluation of hematology and blood chemistry; periodic measurement of vital signs; and the performance of physical examinations, as detailed in the schedule of procedures and assessments of the protocol.

### Follow-up Phase:

Duration of Follow-up Phase is determined based on whether or not subject has experienced virologic failure during the Treatment Extension Phase.

 Subjects receiving PRO 140 350mg and 525mg who experience virologic failure and do not elect to receive the higher dose of PRO 140 525mg or 700mg, respectively and all subjects receiving PRO 140




Name of Sponsor:

CytoDyn, Inc.

### Name of Study Product:

PRO 140 (Humanized monoclonal antibody to CCR5)

Protocol Number: Indication:

PRO 140 \_CD03 Extension Human Immunodeficiency Virus Type-1 (HIV-1) Infection

700mg who experience virologic failure during the Treatment Extension Phase, will be assessed every 4 weeks until the viral suppression is achieved (i.e., plasma HIV-1 RNA levels decline to < 50 copies/mL). Additionally, virologic failure subjects will return to clinic for long-term follow-up at 6 months and at one year from the time of the Virologic Failure (VF) Visit.

 Subjects who do not experience virologic failure at the end of Treatment Extension Phase, will be assessed every 2 weeks for total of 4 weeks.

#### **Duration of Treatment:**

- Screening Phase: up to 3 weeks
- Treatment Extension Phase: weekly treatment injection ± allowed windows
- Follow-up Phase:
  - o Non-Virologic Failure (NVF): 4 weeks
  - o Virologic Failure (VF): Until viral suppression is achieved.
    - Additionally, subjects who experience virologic failure will return to clinic for longterm follow-up at 6 months and at one year from the time of the Virologic Failure Visit.

**Inclusion Criteria:** Potential subjects are required to meet all of the following criteria for enrollment into the study.

- 1. Subjects who have completed 48 weeks of treatment in PRO140 CD03 study.
- 2. Last known Plasma HIV-1 RNA < 50 copies/mL within PRO140 CD03 study.
- 3. Both male and female patients and their partners of childbearing potential must agree to use 2 medically accepted methods of contraception (e.g., barrier contraceptives [male condom, female condom, or diaphragm with a spermicidal gel], hormonal contraceptives [implants, injectables, combination oral contraceptives, transdermal patches, or contraceptive rings], and intrauterine devices) during the course of the study (excluding women who are not of childbearing potential and men who have been sterilized). Females of childbearing potential must have a negative serum pregnancy test at Screening visit and negative urine pregnancy test prior to receiving the first dose of study drug.
- 4. Willing and able to participate in all aspects of the study, including use of SC medication, completion of subjective evaluations, attendance at scheduled clinic visits, and compliance with all protocol requirements as evidenced by providing written informed consent.

Exclusion Criteria: Potential subjects meeting any of the following criteria will be excluded from enrollment.

- 1. Not currently enrolled in PRO140 CD03 study.
- 2. Any active infection or malignancy requiring acute therapy (with the exception of local cutaneous Kaposi's sarcoma).






| Na | me | of | Sp | ons | or: |
|----|----|----|----|-----|-----|

CytoDyn, Inc.

### Name of Study Product:

PRO 140 (Humanized monoclonal antibody to CCR5)

**Protocol Number:** Indication:

PRO 140 CD03 Extension Human Immunodeficiency Virus Type-1 (HIV-1) Infection

- 3. Females who are pregnant, lactating, or breastfeeding, or who plan to become pregnant during the study.
- 4. Subjects weighing < 35kg.
- 5. History of anaphylaxis to any oral or parenteral drugs.
- 6. History of Bleeding Disorder or patients on anti-coagulant therapy (except aspirin).
  - Note: Subjects with well-controlled bleeding disorder while on stable anti-coagulant therapy dose with documented stable INRs can be enrolled as per discretion of the Investigator.
- 7. Any other clinical condition that, in the Investigator's judgment, would potentially compromise study compliance or the ability to evaluate safety/efficacy.

### **Statistical Considerations:**

### Sample Size Determination and Rationale:

Sample size determination is not applicable as only those subjects who are currently enrolled in PRO 140 CD 03 study are allowed to participate in this study.

### **Analysis Populations:**

The Safety population is defined as all subjects who received at least one dose of PRO 140 within the PRO 140 CD03 Extension study. This population will be used for the analysis of safety parameters.

All data collected from the study will be presented as a by-subject listing and also summarized according to the variable type as:

- a. Continuous data summaries will include number of observations, mean, standard deviation, median, and minimum and maximum values
- b. Categorical data summaries will include frequency counts and percentages






# TABLE OF CONTENTS

| STUDY ' | FITLE | 1 |
|---|---|---|
| PROTO | COL SYNOPSIS | 5 |
| TABLE | OF CONTENTS | 10 |
| LIST OF T | ABLES | 15 |
| | IGURES | |
| | ABBREVIATIONS | |
| | ODUCTION | |
| | ATEMENT OF INTENT | |
| | E PROBLEM STATEMENT | |
| 1.3 NA | ME AND DESCRIPTION OF THE INVESTIGATIONAL PRODUCT | 21 |
| 1.4 Su | MMARY OF PRIOR PRE-CLINICAL AND CLINICAL STUDIES | 22 |
| 1.4.1 | Pre-Clinical Studies with PRO 140. | 22 |
| 1.4.2 | Clinical Studies with PRO 140 | 22 |
| 1.4.2.1 | PRO 140 1101 Study | 22 |
| 1.4.2.2 | PRO 140 1102 Study | 22 |
| 1.4.2.3 | PRO 140 1103 Study | 23 |
| 1.4.2.4 | PRO 140 1302 Study | 23 |
| 1.4.2.5 | PRO 140 2301 Study | 26 |
| 1.4.2.6 | PRO 140 2101 Study | 26 |
| 1.4.2.7 | PRO 140 _CD01 Study | 29 |
| 1.4.2.8 | PRO 140 _CD01-Extension Study | 30 |
| 1.4.2.9 | PRO 140 _CD02 Study | 31 |
| 1.4.2.10 | PRO 140 _CD02 _Open Label | 31 |
| 1.4.2.11 | PRO 140 _CD02 Extension Study | 31 |
| 1.4.2.12 | PRO 140 _CD03 Study | 32 |
| 1.5 RA | TIONALE FOR DOSE SELECTION | 35 |
| 1.6 RIS | SKS / BENEFITS ASSESSMENT | 36 |
| 1.6.1 | Risks/Discomfort to Subjects and Precautions to Minimize Risk | 36 |
| 1.6.1.1 | Risks associated with using monotherapy treatment | 36 |
| 1.6.1.2 | Allergic Reaction | 36 |
| 1.6.1.3 | Immune Response | 37 |
| 1.6.1.4 | Pregnancy | 37 |
| 1.6.1.5 | Venipuncture for blood sampling and Subcutaneous injection for Study Drug | |
| | Administration | 37 |





| 1.6.1.6 | Risks related to resumption of viral replication in anatomically privileged compartments | 37 |
|---|---|---|
| 1.6.1.7 | Risks to the Study Personnel and the Environment | |
| 1.6.1.8 | Unknown Risks | |
| 1.6.1.9 | Theoretical risk for increased severity of West Nile virus infection | 37 |
| 1.6.2 | Intended Benefit for Subjects | |
| 2 STUI | OY OBJECTIVES | 39 |
| | OY DESIGN | |
| 3.1 ST | JDY CENTER(S) | 41 |
| 3.2 ST | JDY POPULATION | 41 |
| 3.3 EL | GIBILITY CRITERIA | 41 |
| 3.3.1 | Inclusion Criteria | |
| 3.3.2 | Exclusion Criteria | |
| 4 STUI | OY SCHEDULE | 44 |
| 4.1 Sc. | REENING PHASE | 49 |
| 4.1.1 | Screening Phase | |
| 4.2 TR | EATMENT EXTENSION PHASE | 50 |
| 4.2.1 | Treatment Extension Phase: Treatment Extension Visit-1 (TE1) | 52 |
| 4.2.2 | Treatment Extension Phase: Subsequent Treatment Extension Visits | 53 |
| 4.2.3 | Treatment Extension Phase: End of Treatment Visit (EOT) | 54 |
| 4.3 VII | ROLOGIC FAILURE (VF) VISIT | 55 |
| 4.4 Fo | LLOW-UP PHASE | 56 |
| 4.4.1 | Follow-Up Visits | 57 |
| 4.4.1.1 | Short-Term Follow-Up Visits | 57 |
| 4.4.1.1.1 | Virologic Failure Subjects | 57 |
| 4.4.1.1.2 | Non Virologic Failure Subjects | 57 |
| 4.4.1.2 | Long-Term Follow-Up Visits | 58 |
| 5 SUBJ | ECT COMPLETION AND WITHDRAWAL | 59 |
| 5.1 Su | BJECT COMPLETION | 59 |
| 5.2 Su | BJECT WITHDRAWAL | 59 |
| 5.2.1 | Discontinuation of Study Treatment | 60 |
| 5.2.2 | Data Collected for Withdrawn Subjects | 60 |
| 5.3 SC | reen Failures | 60 |
| 6 STUI | OY TREATMENT | 62 |
| 6.1 Inv | /ESTIGATIONAL PRODUCT DESCRIPTION | 62 |





| 6.2 | INVESTIGATIONAL PRODUCT PACKAGING AND LABELING | 63 |
|-------|-----------------------------------------------------------------|----|
| 6.3 | Investigational Product Storage | 66 |
| 6.4 | INVESTIGATIONAL PRODUCT ADMINISTRATION | 67 |
| 6.5 | INVESTIGATIONAL PRODUCT RECEIPT AND ACCOUNTABILITY | 67 |
| 6.6 | Investigational Product Disposition | 68 |
| 7 D | DESCRIPTION OF PROTOCOL ASSESSMENTS AND PROCEDURES | |
| 7.1 | INFORMED CONSENT | |
| 7.2 | ASSESSMENT OF ELIGIBILITY | |
| 7.2.1 | Re-screening | |
| 7.3 | DEMOGRAPHIC INFORMATION | |
| 7.4 | MEDICAL HISTORY | |
| 7.5 | CONCOMITANT MEDICATIONS AND NON-STUDY TREATMENTS | |
| 7.5.1 | Excluded Medications and Therapies | |
| 7.5.2 | - | |
| 7.6 | PHYSICAL EXAMINATION | 71 |
| 7.7 | Electrocardiogram | 72 |
| 7.8 | NEUROLOGICAL ASSESSMENT | |
| 7.9 | VITAL SIGNS | |
| 7.10 | | |
| 7.10. | | |
| 7.10. | | |
| 7.10. | • | |
| 7.10. | - | |
| 7.10. | 5 Urine pregnancy test | 73 |
| 7.10. | 6 Plasma HIV-1 RNA level and TruCount T Assay | 73 |
| 7.10. | 7 HIV-1 Trofile® DNA Assay | 74 |
| 7.10. | 8 HIV-1 Trofile® RNA Assay | 74 |
| 7.10. | 9 HIV-1 Drug Resistance Assay | 74 |
| 7.10. | 10 Plasma HIV-1 RNA Single Copy Assay | 75 |
| 7.10. | PK sample for PRO 140 | 75 |
| 7.10. | 12 Anti-idiotypic antibodies to PRO 140 | 75 |
| 7.10. | 13 PhenoSense® Entry Assay | 75 |
| 7.10. | 14 CCR5 Receptor Occupancy | 75 |
| 7.10. | 15 All laboratory reports will be reviewed by the Investigator. | 76 |
| 7.11 | PRO 140 Administration | 76 |





| 7.12 | INJECTION SITE REACTION ASSESSMENT | 76 |
|--------|-------------------------------------------|----|
| 7.13 | COVID-19 GUIDANCE | 76 |
| 8 S | TATISTICAL CONSIDERATIONS | 78 |
| 8.1 | Treatment Groups | 78 |
| 8.2 | DESCRIPTION OF STUDY OUTCOME MEASURES | |
| 8.2.1 | Primary Outcome Measures | |
| 8.2.2 | Secondary Outcome Measures | |
| 8.2.3 | Safety Assessments | |
| 8.3 | SAMPLE SIZE DETERMINATION AND RATIONALE | 79 |
| 8.4 | RANDOMIZATION AND BLINDING | 79 |
| 8.5 | Interim Analysis | 79 |
| 8.6 | GENERAL STATISTICAL CONSIDERATIONS | 79 |
| 8.6.1 | Analysis Populations | 79 |
| 8.6.2 | Statistical Methods | 79 |
| 8.6.3 | Prognostic Factors/Covariates | 79 |
| 8.6.4 | Handling of Missing Data | 79 |
| 8.6.5 | Multicenter Study | 79 |
| 8.7 | Data Summary | 79 |
| 8.7.1 | Subject Disposition | 79 |
| 8.7.2 | Demographic and Baseline Characteristics | 80 |
| 8.7.3 | Prior and Concomitant Medications | 80 |
| 8.7.4 | Efficacy Analysis | 80 |
| 8.7.5 | Safety Analysis | 80 |
| 8.7.5. | 1 Adverse Events | 80 |
| 8.7.5. | 2 Tolerability Assessment | 81 |
| 8.7.5. | 3 Clinical Laboratory Data | 81 |
| 8.7.5. | 4 Physical Examination | 81 |
| 8.7.5. | 5 Vital Signs | 81 |
| 8.7.5. | 6 ECG Examination | 81 |
| 8.7.5. | 7 Neurological Assessment | 81 |
| 9 A | DVERSE EVENTS (DEFINITIONS AND REPORTING) | 82 |
| 9.1 | Adverse Event | 82 |
| 9.1.1 | Reporting of Adverse Events | 82 |
| 9.1.2 | Impact of Study Treatment | |
| 9.1.3 | DAIDS AE Grade (Severity) Assessment | |
| 9.1.4 | Causality Assessment | 83 |





| 9.1.5 | Treatment Given as a Result of the Event | 84 |
|---|---|---|
| 9.1.6 | Outcome Assessment | 84 |
| 9.1.7 | Expected / Anticipated Adverse Events | 85 |
| 9.1.8 | SC Injection-related Events | 85 |
| 9.2 | SERIOUS ADVERSE EVENTS (SAE) | 85 |
| 9.2.1 | Reporting of Serious Adverse Events | 86 |
| 9.2.2 | SAE Follow-Up | 87 |
| 10 D | IRECT ACCESS TO SOURCE DATA/DOCUMENTATION | 88 |
| 11 Q | UALITY CONTROL AND QUALITY ASSURANCE | 89 |
| 11.1 | MONITORING REQUIREMENTS | 89 |
| 11.2 | ACCEPTABILITY OF CASE REPORT FORMS (CRFs) | 89 |
| 11.3 | MODIFICATION OF PROTOCOL | 89 |
| 11.4 | REPORTING PROTOCOL DEVIATIONS | 90 |
| 12 E | THICS AND REGULATORY REQUIREMENTS | 91 |
| 12.1 | INSTITUTIONAL REVIEW BOARD/INDEPENDENT ETHICS COMMITTEE (IRB/IEC) | 91 |
| 12.2 | Investigator's Responsibilities | 91 |
| 12.3 | SUBJECT INFORMED CONSENT REQUIREMENTS. | 92 |
| 13 D | ATA HANDLING AND RECORD KEEPING | 93 |
| 13.1 | RECORDING AND COLLECTION OF DATA | 93 |
| 13.2 | CLINICAL DATA MANAGEMENT | 93 |
| 13.3 | Archiving | 93 |
| 14 P | UBLICATION PLAN | 95 |
| 15 R | EFERENCES | 96 |
| 16 A | PPENDIX | 99 |
| 16.1 | APPENDIX I: AIDS-DEFINING CONDITIONS | 99 |
| | APPENDIX II: DIVISION OF AIDS TABLE FOR GRADING THE SEVERITY OF ADULT AND ATRIC ADVERSE EVENTS (DAIDS AE GRADING TABLE) | 101 |
| 16.3 | APPENDIX III: ADVERSE EVENTS OF SPECIAL INTEREST: INJECTION SITE REACTIONS | 102 |
| 16.4 | APPENDIX V: NEUROLOGICAL ASSESSMENT | 103 |





# LIST OF TABLES

| Table 1-1: | Clinical Studies with PRO 140. | 33 |
|---|---|---|
| Table 4-1: | Schedule of Assessments – Screening and Treatment Extension Phase | 45 |
| Table 4-2: | Schedule of Assessments –Follow-Up (FU) Phase | 47 |
| Table 4-3: | Two Groups , Treatment Extension Phase | 50 |
| Table 6-1: | Investigational Product - PRO 140 | 63 |
| Table 9-1: | DAIDS AE Grading General Guidelines | 83 |




# LIST OF FIGURES

| Figure 1-1: | PRO 140 1302 Study: Mean of the maximum (nadir) log <sub>10</sub> reductions in HIV | RNA<br>24 |
|---|---|---|
| Figure 1-2: | PRO 140 1302 Study: Mean log <sub>10</sub> reductions in HIV RNA over time | 24 |
| Figure 1-3: | PRO 140 1302 Study: PRO 140 serum concentrations following a single intravenous injection in HIV- infected individuals. | 25 |
| Figure 1-4: | PRO 140 2301 Study: Mean change from baseline in HIV-1 RNA (Log10 copies/mL) over Time (ITT Subjects) | 26 |
| Figure 1-5: | PRO 140 2101 Study: Mean of the maximum (nadir) log <sub>10</sub> reductions in HIV | RNA<br>27 |
| Figure 1-6: | PRO 140 2101 Study: Mean change from baseline in HIV-1 RNA (Log <sub>10</sub> copies/mL) over Time (ITT Subjects) | 28 |
| Figure 1-7: | Change in CD4+ cell counts in subjects treated with subcutaneous PRO 140 | 28 |
| Figure 1-8: | Emax analysis of antiviral data generated with IV and SC PRO 140 | 35 |
| Figure 3-1: | Study Flow Diagram | 43 |
| Figure 6-1: | PRO 140 (CHO) 175mg/mL - Vial Label | 64 |
| Figure 6-2: | PRO 140 (CHO) 175mg/mL - Syringe Label | 64 |
| Figure 6-3: | PRO 140 (CHO) 175mg/mL - Kit Label | 65 |






# **LIST OF ABBREVIATIONS**

| AE Adverse Event AIDS Acquired Immune Deficiency Syndrome ALT Alanine Transaminase ANC Absolute Neutrophil Count ART Anti Retroviral Therapy AST Aspartate Transaminase ATC Anatomic Therapeutic Classification |
|---|
| ALT Alanine Transaminase ANC Absolute Neutrophil Count ART Anti Retroviral Therapy AST Aspartate Transaminase |
| ANC Absolute Neutrophil Count ART Anti Retroviral Therapy AST Aspartate Transaminase |
| ART Anti Retroviral Therapy AST Aspartate Transaminase |
| AST Aspartate Transaminase |
| ATC Anatomic Therapeutic Classification |
| Indiana Indiapentia Ciassification |
| AUC Area Under Curve |
| °C Celsius |
| cART Combination Antiretroviral Therapy |
| CBC Complete Blood Count |
| CCR5 C-C chemokine receptor type 5 |
| CDC Centers for Disease Control and Prevention |
| CFR Code of Federal Regulations |
| CHO Chinese Hamster Ovary |
| Cm Centimeter |
| CRF Case Report Form |
| C <sub>max</sub> Maximal Concentration |
| CRO Contract Research Organization |
| CS Clinically Significant |
| DAIDS Division of AIDS |
| DMC Data Monitoring Committee |
| DNA Deoxyribonucleic Acid |
| DO Doctor of Osteopathic Medicine |
| ECG Electrocardiogram |
| eCRF Electronic Case Report Form |
| Emax Maximum drug effect |
| et al et aliae; Latin for "and others" |
| °F Fahrenheit |
| FDA U.S. Food and Drug Administration |
| FDP Fixed Dose Procedure |
| FU Follow-Up |
| GCP Good Clinical Practice |
| HAART Highly Active Antiretroviral Therapy |
| Hb Hemoglobin |
| HCT Hematocrit |




| Abbreviation | Term |
|--------------|-------------------------------------------------|
| HEENT | Head, Ears, Eyes, Nose, and Throat |
| HIPAA | Health Insurance Portability Accountability Act |
| HIV | Human Immunodeficiency Virus |
| IA | Interim Analysis |
| IB | Investigator's Brochure |
| ICF | Informed Consent Form |
| ICH | International Conference on Harmonization |
| i.e. | id est; Latin for "that is" |
| IEC | Independent Ethics Committee |
| IND | Investigational New Drug |
| INR | International Normalized Ratio |
| IP | Investigational Product |
| IRB | Institutional Review Board |
| ISR | Injection Site Reactions |
| IV | Intravenous |
| LDH | Lactate dehydrogenase |
| LPN | Licensed Practical Nurse |
| LVN | Licensed Vocational Nurse |
| mAb | Monoclonal Antibody |
| MD | Doctor of Medicine |
| MedDRA | Medical Dictionary for Regulatory Activities |
| Mg | Milligram |
| mL | Milliliter |
| Mm | Millimeter |
| MW | Molecular Weight |
| NCS | Not Clinically Significant |
| NP | Nurse Practitioner |
| NTF | Non-Treatment Failure |
| OBT | Optimized Background Therapy |
| PA | Physician Assistant |
| PI | Principal Investigator |
| PK | Pharmacokinetics |
| PP | Per protocol |
| PT | Prothrombin Time |
| QC | Quality Control |
| RBC | Red Blood Cells |
| RN | Registered Nurse |






| Abbreviation | Term |
|--------------|-----------------------------------|
| RNA | Ribonucleic acid |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SC | Subcutaneous |
| SD | Standard Deviation |
| SOP | Standard Operating Procedure |
| SV | Screening Visit |
| TEAE | Treatment Emergent Adverse Events |
| TF | Treatment Failure |
| USA | United States of America |
| VF | Virologic Failure |
| WBC | White Blood Cells |




#### 1 INTRODUCTION

#### 1.1 STATEMENT OF INTENT

The design, conduct and reporting of this trial shall be conducted in compliance with the protocol, International Conference on Harmonization/Good Clinical Practice (ICH/GCP), and all appropriate regulatory requirements. Investigator(s) participating in this study will have documented training in GCP. Independent monitoring of the trial will be accomplished utilizing as the Contract Research Organization (CRO).

### 1.2 THE PROBLEM STATEMENT

Substantial progress has been made over the past two decades in the development of effective and well tolerated combination antiretroviral regimens. Most HIV-1 infected persons who initiate antiretroviral therapy at early stages in the disease process and who are fully adherent to their antiretroviral regimens can anticipate life expectancies that are measured in decades. Although these advances have revolutionized antiretroviral therapy for most HIV-1 infected patients, contemporary lifelong daily adherence to treatment regimens remains challenging for a significant subset of patients. A number of studies have been conducted to evaluate the possibility of treatment simplification following control of viral replication with an induction regimen [Arribas JR, 2005][Pulido F, 2008][Moltó J, 2007] [Cameron DW, 2008][Nunes EP, 2009][Meynard JL, 2010][Katlama C, 2010][Gutmann C, 2010][Cahn P, 2011][Guiguet M et al., 2012]. Most of these simplification trials have involved the substitution of a boosted HIV-1 protease inhibitor such as lopinavir or darunavir for an effective combination regimen. Although the strategy has been successful in a substantial fraction of those who undergo regimen simplification, the overall body of evidence suggests that boosted protease inhibitor maintenance therapy is generally less effective than maintenance on a three drug regimen [Calza L, 2012][Thompson MA, 2012]. Factors influencing the likelihood of success include the duration of successful suppression prior to the regimen simplification and the extent to which patients are adherent to their simplified regimens [Calza L, 2012]. Although it has also been suggested that some patients may fail because of variability in trough concentrations of protease inhibitors, this has not been substantiated in rigorously conducted studies [Boffito M, 2003]. Other concerns that have been raised include the ability of HIV-1 protease inhibitors to achieve suppressive levels in the central nervous system [Thompson MA, 2012]. The current consensus appears to be that this approach should be reserved for specific patient populations in which considerations related to chronic nucleoside toxicity and/or adherence to complex antiretroviral regimens are dominant. In these situations, the importance of adherence and of close monitoring of plasma HIV-1 RNA levels has been




emphasized. In the case of HIV-1 protease inhibitor maintenance therapy, reestablishment of control of retroviral replication has generally been achieved by resumption of combination therapy.

Also, there is an interest in the development of infrequently administered therapy both as a treatment and a prevention strategy. The Long-Acting Antiretroviral Treatment Enabling (LATTE) study tested a combination of two oral antiretroviral drugs, the non-nucleoside reverse transcriptase inhibitor rilpivirine and the new integrase inhibitor GSK1265744[Spreen WR, 2013]. Furthermore, a long-acting injectable medication can be an effective approach to circumvent the need for daily medication adherence and/or chronic nucleoside toxicity.

Although PRO 140 would require either subcutaneous (SC) or intravenous (IV) administration, its favorable pharmacokinetics might allow dosing as infrequent as once weekly or bi-weekly. The ability to administer the drug infrequently under medical supervision could obviate one of the continuing challenges of close adherence to daily boosted protease inhibitor regimens that appear to be relatively unforgiving in maintenance settings when administered as the sole antiretroviral regimen. This is an open-label study of PRO 140 monotherapy as maintenance therapy for subjects previously fully suppressed on combination antiretroviral regimen. PRO 140 is a promising new antiretroviral agent that does not show any cross-resistance with drugs from other classes. The purpose of this study is to assess the clinical safety and treatment strategy of using PRO 140 SC as long-acting, single-agent maintenance therapy for the chronic suppression of CCR5-tropic HIV-1 infection.

### 1.3 NAME AND DESCRIPTION OF THE INVESTIGATIONAL PRODUCT

PRO 140 is a humanized IgG4,κ monoclonal antibody (mAb) to the C-C chemokine receptor type 5 (CCR5), under development as a therapy for human immunodeficiency virus (HIV) infection.

PRO 140 binds to the N terminus (Nt) and the extracellular loop 2 (ECL2) domain of the CCR5 cell surface receptor that HIV-1 uses to gain entry to a cell. PRO 140 binding to CCR5 blocks the final phase of viral binding to the cell surface prior to fusion of the viral and cell membranes. PRO 140 has been administered intravenously or subcutaneously to 174 HIV-1 infected individuals in Phase I/II studies of safety, tolerability, pharmacokinetics and pharmacodynamics [Jacobson JM, 2010][Jacobson JM, 2010]. The drug has been well tolerated following administration of single doses of 0.5 to 5 mg/kg or up to three weekly doses of up to 324 mg. Single subcutaneous doses of 324 mg have resulted in drops in plasma HIV-1 RNA levels of approximately 1.0 log<sub>10</sub>. Repetitive weekly administration of this dose of PRO 140 has been associated with drops in plasma HIV-1 RNA levels of approximately 1.5 log<sub>10</sub>. Serum concentrations of PRO 140 above the IC<sub>50</sub> for clinical isolates of HIV-1 are maintained for at least 2 weeks following a single dose of 324 mg. Plasma HIV-1 RNA levels rise to baseline levels as PRO 140 is cleared from the plasma and, presumably, other compartments.




### 1.4 SUMMARY OF PRIOR PRE-CLINICAL AND CLINICAL STUDIES

### 1.4.1 Pre-Clinical Studies with PRO 140

*In vitro* and *in vivo* preclinical studies have been conducted to determine the pharmacokinetic, immunogenicity, and toxicity profiles of PRO 140 following IV and SC administration. Several acute and chronic toxicity studies have been conducted to support the clinical development plan.

Acute toxicity of PRO 140 was evaluated in New Zealand rabbits, following IV administration of 5 or 15 mg/kg. Chronic toxicity was evaluated in cynomolgus monkeys following biweekly administration of IV doses up to 10 mg/kg for six months and biweekly administration of various SC doses up to 50 mg/kg for 24 weeks. The drug was generally well tolerated. Biweekly administration of IV doses up to 10 mg/kg for six months resulted in minimum to mild lymphoid hyperplasia in assorted lymph nodes and spleen, which was considered an expected immune response to a foreign protein. Biweekly administration of SC doses up to 50 mg/kg for 24 weeks resulted in minimum injection-site reactions (minimal, multifocal, mononuclear cell infiltrates in the subcutis), which were considered due to an inflammatory response to the injected antigen. Monkeys tolerated treatment with PRO 140 for 24 weeks without evidence of local or systemic toxicity. PRO 140 caused no mortality, cageside observations, in-life injection-site observations, or gross pathologic findings. Chronic treatment with PRO 140 did not affect body weight, food consumption, hematology, clinical chemistry or coagulation parameters.

Both IV and SC administration resulted in elimination half-lives of approximately 200 hours, and overall exposure increased with increasing doses. Following SC administration of PRO 140 in monkeys, the maximal concentration ( $C_{max}$ ) was achieved within 56 hours and bioavailability for PRO 140 after SC dosing was approximately 70%.

### 1.4.2 Clinical Studies with PRO 140

Current human experience with PRO 140 consists of seven completed and two ongoing clinical trials. These studies are summarized in Table 1-1. In all the completed clinical trials, the majority of adverse events (AEs) were mild or moderate. No dose-limiting toxicities or patterns of drug-related toxicities were observed. Antiviral activity was potent, rapid, prolonged, dose-dependent, and highly significant.

### 1.4.2.1 PRO 140 1101 Study

For the first-in-human trial, PRO 140 1101, the drug was administered IV at 0.1, 0.5, 2.0, or 5.0 mg/kg and was generally well tolerated, non-immunogenic, and without clinically relevant toxicity. Treatment Emergent Adverse Events (TEAEs) did not increase with rising PRO 140 dose levels. 75% of subjects reported TEAEs, most of which were deemed unrelated to study treatment.

### 1.4.2.2 PRO 140 1102 Study




In PRO 140 1102 study, the majority of AEs, other than injection-site reactions, were considered mild and possibly related to drug administration. The majority of injection-site reactions were considered mild, self-resolving, and definitely related to drug administration. PRO 140 derived from Chinese Hamster Ovary (CHO) cells and administered SC at 100 mg/mL was generally well tolerated in healthy, normal volunteers. Overall, PRO 140 administered SC using Autoject® 2 appeared better tolerated than manual injection.

# 1.4.2.3 PRO 140 1103 Study

In PRO 140 1103 study, administration of PRO 140 at 350 mg using Autoject® 2 appeared well tolerated. Manual injections, on the other hand, were associated with a greater number of AEs. There did not appear, however, to be any substantial difference in subject perception of pain or discomfort related to site of drug administration. No anti-PRO 140 antibodies were detected in any subjects in this study. There was a tendency of higher exposure associated with SC administration of PRO 140 at 350 mg in the abdomen and the thigh. A higher number of AEs was associated with injections in the arm. Based on these observations, thigh and abdominal administration of PRO 140 were preferred over arm injection.

### 1.4.2.4 PRO 140 1302 Study

This initial proof-of-concept study was a randomized, double-blind, placebo-controlled study in subjects with early-stage, asymptomatic HIV infection, only R5 HIV-1 detectable, and no antiretroviral therapy for 12 weeks. Subjects (n=39) were randomized to receive a single IV injection of placebo or PRO 140 at doses of 0.5, 2, or 5 mg/kg. Subjects were monitored for antiviral effects, safety and PRO 140 pharmacokinetics (PK) for 58 days.

The study enrolled 31 males and 8 females. The median age,  $CD4^+$  cell count and HIV-1 RNA at baseline were 40.3 years, 484cells/ $\mu$ L and 26,900 copies/mL, respectively. The baseline characteristics were similar for all treatment groups.

PRO 140 demonstrated potent, rapid, prolonged and dose-dependent antiviral activity (Figure 1-1 and Figure 1-2). A single 5mg/kg dose reduced viral loads by 1.83 log<sub>10</sub> on average (Figure 1-2). These reductions represent the largest antiviral effects reported after just one dose of any HIV-1 drug [Jacobson JM, 2008]. In the 5 mg/kg group, mean viral load reductions of greater than 1 log<sub>10</sub> were sustained for 2-3 weeks post-treatment (Figure 1-2).




Figure 1-1: PRO 140 1302 Study: Mean of the maximum (nadir) log<sub>10</sub> reductions in HIV RNA



Figure 1-2: PRO 140 1302 Study: Mean log<sub>10</sub> reductions in HIV RNA over time



There was no change in R5 virus susceptibility to PRO 140 following treatment. All subjects had R5-only virus at screening in the first-generation Trofile assay. R5-only tropism results were observed in all subjects at all other time points, with two exceptions: One of nine (11%) of placebo subjects had dual/mixed virus at baseline and all subsequent time points, reflecting a spontaneous




and stable switch in co-receptor tropism results. One of 30 (3%, 0.5 mg/kg group) had a dual/mixed tropism result on day 8 and R5-only results at all other time points, including the end of the day [Jacobson JM, 2008]. Clonal analysis of the dual/mixed virus revealed that it reflected outgrowth of pre-existing undetected virus rather than mutation of an R5 virus to a dual/mixed virus following treatment [Marozsan, 2008]. Therefore, no significant development of viral resistance to PRO 140 was observed despite potent and prolonged (2-3 weeks on average) viral suppression, followed by slow washout of the drug. Given that resistance to other classes of HIV-1 drugs can develop within one week of monotherapy [Demeter LM, 2000] [Saag, 1993][Richman, 1994], the findings indicate that PRO 140 presents a high barrier to viral resistance in vivo.

Figure 1-3 illustrates the mean serum concentrations of PRO 140 after IV injection. Serum levels increased with increasing dose. The mean Area Under Curve (AUC) from time zero to infinity (AUC∞) values were 11.1, 74.3 and 278 mg x day/L for the 0.5, 2 and 5 mg/kg groups. The mean serum half-life was 3.5-3.9 days in the two highest dose groups. In addition, PRO 140 significantly masked CCR5 on circulating lymphocytes for 2-4 weeks [Jacobson JM, 2008]. The PK and receptor occupancy data were broadly consistent with the duration of antiviral effects.

Figure 1-3: PRO 140 1302 Study: PRO 140 serum concentrations following a single intravenous injection in HIV- infected individuals.



The figure illustrates the mean serum concentrations over time by treatment group. The error bars depict standard deviations. The mean serum half-lives were 3.9 days and 3.5 days in the 2 mg/kg and 5 mg/kg dose groups, respectively.

Intravenous PRO 140 was generally well tolerated. No drug-related serious events or dose-limiting toxicity was observed. The most common adverse events (headache, lymphadenopathy, diarrhea, and fatigue) were observed at similar frequencies across the placebo and PRO 140 dose groups.




There was no significant effect on QTc interval intervals or other electrocardiographic parameters, and there were no remarkably laboratory findings. There was no loss or depletion of CD4<sup>+</sup> or CCR5<sup>+</sup> cells from the circulation. At the 5 mg/kg dose, there was a trend towards increased CD4<sup>+</sup> cell counts from baseline, with mean changes of +129, +96 and +83 cells/μL observed on days 8, 15, and 22, respectively.

# 1.4.2.5 PRO 140 2301 Study

PRO 140 2301 was a multi-center, randomized, double-blind, placebo-controlled, parallel group study in 30 male and female adult subjects infected with HIV-1. Subjects were randomized to one of three groups (N=10/group), each receiving one of three treatments: (i) a single IV dose of 5 mg/kg by 30-minute IV infusion; (ii) a single IV dose of 10 mg/kg by 30-minute IV infusion; (iii) a single placebo dose by 30-minute IV infusion. The objective of the study was to assess and characterize the PK and PD of PRO 140 administered by IV infusion, assess efficacy at a new dosage level, and safety and tolerability of single doses of PRO 140.

All PRO 140-treated subjects had more than 10-fold reduction in viral loads (mean max log10 reductions were 1.83 for treatment groups and 0.32 for placebo) (Figure 1-4). Both the 5 mg/kg and 10 mg/kg doses have shown favorable tolerability and no dose-limiting toxicity has been observed. High levels of receptor occupancy (> 85% reduction in the number of cells detected) were observed for 29 days after treatment with both 5 and 10 mg/kg doses.

Figure 1-4: PRO 140 2301 Study: Mean change from baseline in HIV-1 RNA (Log10 copies/mL) over Time (ITT Subjects)



# 1.4.2.6 PRO 140 2101 Study






A subcutaneous (SC) form of PRO 140 was tested in HIV-infected subjects. The trial was a randomized, double-blind, placebo-controlled study in subjects (n=44) with early-stage, asymptomatic HIV infection, only R5 HIV-1 detectable, and no antiretroviral therapy for 12 weeks [Thompson, 2009]. Placebo (n=10) and three PRO 140 doses were examined: 162mg weekly for three weeks (n=11), 324mg weekly for three weeks (n=11), and 324mg biweekly (every other week) for two doses (n=12). Subjects were followed for 44 days after the final dose. The study enrolled 40 males and 4 females. The median age, weight, CD4<sup>+</sup> cell count and HIV-1 RNA at baseline were 42.3 years, 79.1 kg, 410 cells/μL and 20,000 copies/mL, respectively. Baseline characteristics were similar for the different treatment groups.

Potent, dose-dependent and highly statistically significant antiviral activity was observed (Figure 1-5 and Figure 1-6). The 324mg weekly dose resulted in a mean 1.65 log<sub>10</sub> reduction in viral load, and highly significant reductions were observed for the other dose groups as well (Figure 1-5). There was no viral rebound between 324mg doses, and the antiviral effects persisted for one week after the final dose Figure 1-6. The trial established the first antiviral proof of concept for a long-acting, self-administrable drug for HIV-1 infection [Thompson, 2009].

Figure 1-5: PRO 140 2101 Study: Mean of the maximum (nadir) log<sub>10</sub> reductions in HIV RNA








Figure 1-6: PRO 140 2101 Study: Mean change from baseline in HIV-1 RNA (Log<sub>10</sub> copies/mL) over Time (ITT Subjects)



Subcutaneous PRO 140 was generally well tolerated both locally and systemically. There was no obvious dose-related pattern of toxicity. The most common adverse events (diarrhea, headache, lymphadenopathy and hypertension) were mild to moderate and self-resolving. These events are common in HIV infection and were reported with similar frequencies in the placebo and PRO 140 treatment groups. Administration-site reactions were mild, transient, and observed in a fraction of subjects. There was a trend towards increased CD4+ cell counts in subjects treated with PRO 140 (Figure 1-7). Based on its encouraging antiviral and tolerability profiles and the convenience of weekly self-administration, SC PRO 140 has been selected for further clinical development.

Figure 1-7: Change in CD4+ cell counts in subjects treated with subcutaneous PRO 140.

Subjects (n=10 to 12 per group) were randomized to received placebo weekly (Days 1, 8, 15), 162mg PRO 140 weekly (Days 1, 8, 15), 324mg PRO 140 biweekly (Days 1, 15, with placebo on Day 8), or 324mg PRO 140 weekly (Days 1, 8, 15). CD4+ cell counts were measured over time, and the median change from baseline was determined for each treatment group.








# 1.4.2.7 PRO 140 CD01 Study

PRO 140 CD01 study (open-label, 43 subjects, multi-center) (12-cohort 1, 28-cohort 2, 3-cohort 3) evaluated the efficacy, safety, and tolerability of PRO 140 monotherapy (350 mg subcutaneous injection weekly for up to 12 weeks) for the maintenance of viral suppression following substitution of antiretroviral therapy in HIV-1 infected patients (with exclusive CCR5-tropic virus). Participants in this study were experienced HIV-infected individuals who were virologically suppressed on combination antiretroviral therapy. Consenting patients were shifted from combination antiretroviral regimen to PRO 140 monotherapy for 12 weeks.

Forty (43) subjects (M/F: 40/3) with median age of 55 years (26-72) and median CD4 T-cell count of 604.5 cells/mm3 (365-1240) were enrolled in the CD01 study. Overall, twenty-three out of 43 (54%) enrolled subjects completed 12 weeks of PRO140 monotherapy without experiencing virologic failure. Virologic failure was defined as two consecutive HIV-1 RNA levels of  $\geq 400$ copies/mL separated by at least 3 days.

Of the first 40 enrolled subjects enrolled under cohort 1 and cohort 2, three subjects were found to have Dual/Mixed (D/M) tropism [1 at baseline and 2 at the time of virologic failure] and 37 subjects were found to have exclusive CCR5-tropic virus. A letter of amendment was filed to




increase the planned number of subjects from 40 to 43 subjects to compensate for the 3 Dual/Mixed subjects enrolled in the study.

All virologic failure subjects who had available lab data in both studies achieved viral suppression to < 400 HIV-1 RNA copies/mL, as well as viral suppression to 'Non Detectable' or < 50 HIV-1 RNA copies/mL after re-initiation of ART.

The by-subject analysis of PhenoSense<sup>®</sup> Entry Assay data for PRO140, maraviroc, and AMD3100 shows no significant changes in the post-treatment IC<sub>50</sub> and IC<sub>90</sub> values were noted when compared with baseline values in virologic failure and non-virologic failure groups of subjects.

Anti-PRO140 antibodies were not identified in any post-treatment sample and data derived from the CD01 study further supports the favorable PRO140 PK profile data generated from both preclinical as well as prior Phase 1/2 clinical trials.

Safety data were analyzed for all 43 enrolled subjects. One (1) of 43 subjects experienced an SAE that was deemed not related to the study drug by the Principal Investigator. Twenty-nine (29) of 43 subjects (67%) experienced one or more adverse events (AEs) after receiving at least one dose of PRO140. The most commonly occurring AEs were infections and infestation conditions which were reported by 14 of 43 (32.5%) subjects. The majority of the reported AEs (62/87; 71.2%) were deemed either unlikely or not related to study treatment by the Investigator. Similarly, the majority of the reported AEs (70/87; 80.4%) were deemed mild in nature.

# 1.4.2.8 PRO 140 CD01-Extension Study

PRO 140\_CD01-Extension study (open-label, 17 subjects, multi-center) seeks to evaluate the efficacy, safety, and tolerability of PRO 140 monotherapy (350 mg subcutaneous injection weekly for up to 160 weeks) for the continued maintenance of viral suppression following substitution of antiretroviral therapy in HIV patients (with exclusive CCR5-tropic virus). Participants in this study were HIV-infected individuals who were virologically suppressed on combination antiretroviral therapy and completed the first 12 weeks of CD01 study without experiencing virologic failure. As with the CD01 study, virologic failure was defined as two consecutive HIV-1 RNA levels of ≥ 400 copies/mL separated by at least 3 days. Consenting patients may remain on PRO 140 monotherapy for up to 160 weeks.

A total of 17 subjects participated in the CD01-Extension study of which one subject was considered not eligible as subject experienced virologic failure prior to first extension treatment.

Sixteen (16) eligible subjects (M/F: 14/2) with median age of 54.9 years (26-68) and median CD4 T-cell count of 593 cells/mm3 (365-1059) were enrolled in an extension study. One patient discontinued at week 37 (with viral load of <40 copies/mL) due to relocation. Two subjects were withdrawn due to non-treatment related SAEs at week 140 and 149, respectively. One subject was withdrawn due to re-starting their ART at week 99. Two subjects withdrew consent at week 81 and 139, respectively. Five (5) subjects experienced virologic failure (VF) (two consecutive viral




load of ≥400 copies/mL). The mean time to virologic failure was 329 days (106-691).

Five (5) subjects are currently receiving weekly 350 mg PRO140 SC monotherapy and have completed more than three years of treatment (176-198 weeks). Overall, 12 subjects completed at least one year of treatment and 9 subjects completed at least two years of treatment in this study.

PRO 140 was generally well tolerated, and no drug-related SAEs were observed.

The clinical study is currently ongoing.

# 1.4.2.9 PRO 140 \_CD02 Study

PRO 140\_CD02 study (double blind, placebo controlled, 50 subjects, multi-center) evaluated the efficacy, safety, and tolerability of PRO 140 in combination with existing ART (failing regimen) for one week and Optimized Background Therapy (OBT) for 24 weeks in patients infected with HIV-1. The study population included 50 treatment-experienced HIV-infected adult patients with CCR5-tropic virus who demonstrated evidence of HIV-1 replication despite ongoing antiretroviral therapy with documented history of genotypic or phenotypic resistance to at least one ART drug within three drug classes (or within two or more drug classes with limited treatment options). The options may be limited as a result of drug antiviral class cross-resistance or documented treatment intolerance.

In double-blind treatment period, virally non-suppressed subjects were randomized and treated with either PRO 140 or Placebo in combination with the failing ART regimen for 7 days. The primary efficacy endpoint was proportion of participants with  $\geq 0.5 \log_{10}$  reduction in HIV-1 RNA viral load from baseline at the end of the 7 day functional monotherapy period.

During the 24-week open-label period, all subjects received PRO 140 along with Optimized Background Therapy (OBT).

This clinical study is completed.

# 1.4.2.10 PRO 140 CD02 Open Label

PRO 140\_CD02\_Open Label (open label, single arm, 25 subjects, multicenter) seeks to evaluate the efficacy, clinical safety, and tolerability parameters of PRO140 in combination with existing ART (failing regimen) for one week and Optimized Background Therapy (OBT) for 24 weeks. The patient population for this trial are treatment-experienced HIV-infected patients with CCR5-tropic virus and demonstrate evidence of HIV-1 replication despite ongoing antiretroviral therapy with documented genotypic or phenotypic resistance to ART drugs within three drug classes (or within two drug classes with limited treatment options).

This clinical study is currently ongoing.

# 1.4.2.11 PRO 140 CD02 Extension Study

PRO 140\_CD02 Extension study (open label, 50 subjects, multi-center) seeks to evaluate the long




term efficacy, safety and tolerability of PRO 140 weekly injection in combination with Optimized Background Therapy (OBT) in patients infected with HIV-1. The study population includes 50 treatment-experienced HIV-infected adult patients with CCR5-tropic virus who successfully completed PRO 140\_CD02 or PRO 140\_CD02\_Open Label study and continue to demonstrate HIV-1 viral suppression.

This clinical study is currently ongoing.

# 1.4.2.12 PRO 140 CD03 Study

PRO 140\_CD03 study (open-label, two-arm comparator, 500 subjects, multi-center) seeks to evaluate the clinical safety and treatment strategy of using PRO 140 SC as a long-acting, single-agent maintenance therapy for 48 weeks in virologically suppressed subjects with CCR5-tropic HIV-1 infection.

The first ~150 eligible subjects were enrolled to receive PRO140 350mg SC weekly injection in a single-arm study. Subsequently, the next ~150 subjects were randomized 1:1 to PRO140 350mg (Group A) or PRO 140 525mg (Group B).

An additional  $\sim$ 200 subjects will be randomized 1:1 to PRO 140 525mg (Group B) or PRO 140 700mg (Group C).

This clinical study is currently ongoing.






**Table 1-1: Clinical Studies with PRO 140** 

| Protocol Number | Phase | No. of<br>Subjects<br>(Planned/<br>Analyzed) | Doses | Cell line used<br>to make PRO-<br>140 | Subject<br>Population | Comments |
|---|---|---|---|---|---|---|
| PRO 140 1101 | 1 | 20/20 | Single 0.1, 0.5, 2.0, or 5.0 mg/kg | Sp2/0<br>myeloma | Healthy | Generally well tolerated; non-immunogenic; dose-<br>dependent coating of CCR5; significant coating of<br>CCR5 over placebo at 0.5, 2, and 5 mg/kg |
| PRO 140 1102 | 1 | 20/20 | Either two or three doses totaling<br>200 or 350 mg respectively | СНО | Healthy | Generally well tolerated; drug derived from CHO cells well tolerated also; SC administration by Autoject® 2 better tolerated than manual injection |
| PRO 140 1103 | 1 | 15/14 | Two doses, each of 350 mg | СНО | Healthy | More AEs associated with arm injection; trend of lower exposure in arm injections; thigh and abdominal administration preferred |
| PRO 140 1302 | 1b | 40/39 | Single 0.5, 2.0, or 5.0 mg/kg | Sp2/0<br>myeloma | HIV-1<br>positive | Generally well tolerated; antiviral suppression<br>maintained for approx. 10 days with higher doses;<br>favorable tolerability and potent, dose-dependent<br>antiviral activity provide proof-of-concept |
| PRO 140 2301 | 2a | 30/31 | Single 5.0 or 10.0 mg/kg | СНО | HIV-1<br>positive | Generally well tolerated with no dose-limiting toxicities; potent antiviral suppression maintained for approx. 20 days when administered IV at 5 or 10 mg/kg. No dose-limiting toxicities at 10 mg/kg. |
| PRO 140 2101 | 2a | 40/44 | Three doses of 162 or 324 mg<br>each | СНО | HIV-1<br>positive | Generally well tolerated, no drug-related SAEs or dose-limiting toxicity; antiviral activity was statistically significant; two-fold exposure at higher dose; single dose demonstrated favorable tolerability, and potent, long-acting, dose-dependent antiviral activity. |
| PRO 140 _CD01 | 2b | 43/43 | 350 mg SC weekly dose for 12<br>weeks of Monotherapy (total<br>treatment duration 14 weeks) | СНО | HIV-1<br>positive | Generally well tolerated, no drug-related SAEs, weekly dose demonstrated favorable tolerability, and potent, long-acting, dose-dependent antiviral activity. Results are pending publication. |




| • | CytoDyn |
|---|---------|
| Щ | СуюДуп |

| PRO 140 _CD01-<br>Extension | 2b | 17/17 | 350 mg SC weekly dose for 160 weeks of Monotherapy (total treatment duration 161 weeks) | СНО | HIV-1 positive | This clinical study is currently ongoing. |
|---|---|---|---|---|---|---|
| PRO 140<br>_CD02 | 2b/3 | 50/52 | Placebo or 350mg SC for 1 dose,<br>followed by 350mg SC weekly<br>dose for 24 weeks (total treatment<br>duration 25 weeks) | СНО | HIV-1<br>positive | This clinical study is completed |
| PRO 140 _CD02_Open Label | 2b/3 | 25/2 | 700mg SC + existing ART for 1<br>week followed by 700mg SC<br>weekly OBT for 24 weeks | СНО | HIV-1 positive | This clinical study is currently ongoing |
| PRO 140 _CD02 Extension | 2b/3 | 50/TBD | 700 mg SC weekly dose in combination with Optimized Background Therapy (OBT) | СНО | HIV-1<br>positive | This clinical study is currently ongoing. |
| PRO 140<br>_CD03 | 2b/3 | 500/TBD | 350 mg, 525 mg, or 700 mg SC<br>weekly dose for 48 weeks of<br>Monotherapy | СНО | HIV-1<br>positive | This clinical study is currently ongoing. |




### 1.5 RATIONALE FOR DOSE SELECTION

The dose of 350 mg administered SC was chosen in light of a previous analysis suggesting that such a dose would be likely to provide maximal viral load suppression.

In studies with antiviral agents that block viral entry through the CCR5 receptor, there is a general consensus that in order to achieve robust antiviral effects and minimize the potential for drug resistance in combination therapy, the dose of drug should result in exposures that fall on the plateau of a Maximum Drug Effect ( $E_{max}$ ) plot.

Figure 1-8: E<sub>max</sub> analysis of antiviral data generated with IV and SC PRO 140.



The maximal viral load reduction was analyzed with regard to drug exposure for PRO 140. Figure 1-8 above shows this relationship. Analysis shows that PRO 140 350mg weekly dose is expected to fall on the plateau of the  $E_{max}$  plot.

The maximal change in HIV-1 viral load from baseline was determined at any point 59 days after initiation of therapy. To allow approximate comparisons between the IV and SC doses, the overall AUC observed for repeat SC doses was conservatively estimated by multiplying the measured AUC<sub>0-7d</sub> by the number of doses administered. Viral load and AUC data were fit to an  $E_{max}$  equation:  $E = E_{max} \times AUC/(AUC + AUC_{50})$ . The orange diamond indicates projected data for three weekly 350 mg doses based on the mean exposure observed in the PRO 140 1103 study.

It is important to note that when larger proteins (MW > 10,000) are administered SC, they initially traffic through the lymphatic system. Uptake into the bloodstream occurs after the proteins reach






the thoracic duct [Nishikawa M, 2005]. In addition, based on pharmacodynamic data from our prior SC and IV studies, maximum virologic suppression is expected to be achieved with trough concentrations that equal or exceed approximately 5  $\mu$ g/mL.

Finally, the mean nadir reduction in viral load achieved with 3 weekly 324 mg SC doses (1.65 log<sub>10</sub>) was similar to the mean nadir reductions observed with single 5 or 10 mg/kg IV doses (1.8 log<sub>10</sub> in each case), and higher viral load reductions are expected in the present study based on the use of the 350 mg CHO formulation. Overall, several lines of evidence indicate that maximum virologic suppression will be achieved with 350 mg weekly dosing in the present study.

Majority of subjects receiving 350 mg weekly SC dosing in monotherapy setting experienced virologic failure in CD01-Extension study. Review of PRO 140 clinical data to date with 350mg SC weekly dosing, suggests no evidence of emergence of viral isolates with reduced susceptibility to PRO 140, no altered viral tropism or anti-PRO 140 antibodies formation suggesting the most likely cause of viral rebound is inadequate dosing to fully cover CCR5 receptor populations. Based on pharmacologic modeling studies, we anticipate that the 525mg and 700 mg dose will result in a lower fraction of study participants with trough levels below that which will 'uncoat' a significant number of CD4 cells (i.e., less than a certain multiple of the IC50 or IC90 for PRO 140).

# 1.6 RISKS / BENEFITS ASSESSMENT

# 1.6.1 Risks/Discomfort to Subjects and Precautions to Minimize Risk

# 1.6.1.1 Risks associated with using monotherapy treatment

Study treatment (PRO 140 350mg, 525mg, or 700 mg SC injection) may not be effective in achieving a reduction in viral load for all subjects. Such cases could lead to an increased risk of developing drug resistance, opportunistic infections and clinical progression of the disease. As patients will not be receiving concomitant antiretroviral drugs of other antiviral classes, should PRO 140 therapy fail, selection of viral variants with reduced susceptibility to these agents would be unlikely (and was not observed in the PRO 140 CD 01 or PRO 140 CD 01-Extension studies).

# 1.6.1.2 Allergic Reaction

PRO 140 belongs to the monoclonal antibody class of drugs. Monoclonal antibodies are sometimes associated with allergic reactions (fatigue, diarrhea, fever, vomiting, headache, nausea, pain at the site of injection, low blood pressure, rash, itching, and chills) or flu-like reactions such as fever, chills, and aches. These events are usually of short duration if they occur at all. Severe allergic reactions, however, can be life-threatening. Although anaphylaxis has not been observed in prior trials of PRO 140, infusion of proteins always carries with it the theoretical risk for anaphylactic shock. Accordingly, whenever PRO 140 is initially administered to subjects, there should be available and in place the procedures required to manage anaphylactic shock.



### 1.6.1.3 Immune Response

Subjects who take PRO 140 or other monoclonal antibodies can also develop an immune response to PRO 140 that may affect their ability to receive monoclonal antibodies, or to benefit from diagnosis or therapy with a monoclonal antibody in the future.

# 1.6.1.4 Pregnancy

Risks to unborn babies are unknown at this time; pregnant females will be excluded from this study. Females of childbearing potential must have a negative pregnancy test prior to enrollment. Both male and female patients and their partners of childbearing potential must agree to use appropriate birth control methods throughout the study duration (excluding women who are not of childbearing potential and men who have been sterilized).

# 1.6.1.5 Venipuncture for blood sampling and Subcutaneous injection for Study Drug Administration

Venipuncture for blood sample collection and subcutaneous injection for study drug administration carries a minimal risk of minor discomfort and the possibility of minor bruising at the site of the needle puncture and, rarely, the possibility of infection at the needle puncture site.

# 1.6.1.6 Risks related to resumption of viral replication in anatomically privileged compartments

It is possible that penetration of PRO 140 into certain key anatomic compartments such as the central nervous system (CNS) or the male genital tract will be insufficient to control viral replication in those locations. Loss of control of viral replication in the CNS could result in the development or exacerbation of HIV-1 Associated Neurocognitive Disorders (HAND) and that a lack of control of HIV-1 replication in the male genital tract could be associated with an increased risk of HIV-1 transmission following unprotected sexual encounters.

# 1.6.1.7 Risks to the Study Personnel and the Environment

The principal risk in the clinical setting is in the handling of needles that may be contaminated with HIV, or other human pathogens. Adherence to universal precautions for working with infectious agents will reduce the risk of exposure to these individuals. All bio-hazardous waste will be disposed of as stipulated by local, state, and federal regulations and in accordance with study site Standard Operating Procedures (SOPs).

### 1.6.1.8 Unknown Risks

As with all research there is the remote possibility of risks that are unknown or that cannot be foreseen based on current information.

# 1.6.1.9 Theoretical risk for increased severity of West Nile virus infection





Individuals who lack a functional CCR5 gene are at increased risk for severe infection by West Nile virus [Thompson, 2009] Because of this, treatment with CCR5 co-receptor antagonists poses a theoretical risk for increased severity of West Nile virus infection. However, this concern is mitigated by several factors. First, no increased risk was observed for individuals who possess one functional and one non-functional CCR5 gene, indicating that an intermediate amount of CCR5 is sufficient for defense against West Nile virus [Thompson, 2009]. Second, use of CCR5 co-receptor antagonists is unlikely to completely abrogate CCR5 function, and there has been no association reported to date between CCR5 co-receptor use and severe West Nile virus. Additionally, PRO 140 weakly antagonizes the natural activity of CCR5 and thus is less likely to adversely affect immune function. Furthermore, this has not been established to be a risk with maraviroc, the anti-CCR5 drug already FDA-approved for the treatment of HIV.

Collectively, the experience with both IV and SC, simulation modeling and the recent confirmation that a higher concentration of PRO 140 synthesized using a highly efficient CHO cell line can be conveniently and safely administered has resulted in the design of the current study.

#### 1.6.2 **Intended Benefit for Subjects**

This study provides an opportunity for subjects to receive once weekly SC treatment with PRO 140. Subjects participating in this Extension monotherapy study will contribute to the development of a drug which has the potential to become a treatment option for them and others in the future.



#### 2 STUDY OBJECTIVES

The objective of this study is to assess the long term safety of using PRO 140 SC as single-agent maintenance therapy for the chronic suppression of CCR5-tropic HIV-1 infection.

The primary outcome measures will be to assess the clinical safety of PRO 140 monotherapy regimen and proportion of participants experiencing virologic failure for all subjects and within each treatment group.

In addition, time to virologic failure for all subjects and within each treatment group, proportion of participants achieving viral re-suppression (HIV-1 RNA < 50 copies/mL) after experiencing virologic failure for all subjects and within each treatment group, time to achieving viral resuppression (HIV-1 RNA < 50 copies/mL) after experiencing virologic failure for all subjects and within each treatment group, proportion of virologic failure subjects achieving viral re-suppression with re-initiation of previous baseline antiretroviral regimen for all subjects and within each treatment group, mean change in CD4 cell count, at each visit within the Treatment Phase for all subjects and within each treatment group.

**Note:** Virologic failure is defined as two (2) consecutive plasma HIV-1 RNA levels of  $\geq 200$  copies/mL.

Safety assessments include evaluation of tolerability of repeated subcutaneous administration of PRO 140 as assessed by investigator –evaluation of injection site reactions for all subjects and within each treatment group, frequency of Grade 3 or 4 adverse events as defined by the DAIDS Adverse Event scale and frequency of treatment-emergent serious adverse events.




3 STUDY DESIGN

This study is an extension study designed to assess the long-term safety of using PRO 140 350mg, 525mg, or 700mg SC as single-agent maintenance therapy for the chronic suppression of CCR5-tropic HIV-1 infection after initial 48 weeks in virologically suppressed subjects.

Consenting subjects will continue weekly PRO 140 350mg, 525mg, or 700mg monotherapy during the Treatment Extension Phase with the one week overlap of existing retroviral regimen and PRO 140 at the end of PRO 140 treatment in subjects who do not experience virologic failure.

Note: Subjects who intend and consent to participate in Treatment Extension phase study will not initiate ART Regimen therapy at T47.

Three groups of subjects included in the study:

- Subjects who continue receiving PRO 140 350mg SC weekly injection
- Subjects who continue receiving PRO 140 525mg SC weekly injection
- Subjects who continue receiving PRO 140 700mg SC weekly injection

Subjects receiving PRO 140 350mg that experience virologic failure during the Treatment Extension phase will have the option of receiving the higher dose of PRO 140 525mg for the remainder of the Treatment Extension phase or may re-initiate prior ART regimen (or an alternative regimen selected by their treating physician).

Subjects receiving PRO 140 525mg that experience virologic failure during the Treatment Extension phase will have the option of receiving the higher dose of PRO 140 700mg for the remainder of the Treatment Extension phase or may re-initiate prior ART regimen (or an alternative regimen selected by their treating physician).

Subjects who move to the higher dose after experiencing virologic failure will continue on treatment at the higher dose from the remaining of the treatment phase. The decision to stop treatment at the higher dose will be at the investigator's discretion based on the subject's viral load at the time of virologic failure, and viral load at subsequent higher dose treatment visits. The study will have three phases: Screening Phase, Treatment Extension Phase and Follow-up Phase.

Screening Phase begins with signing of Informed Consent and lasts up to 21 days. All subjects will continue receiving PRO 140 350mg, 525mg, or 700mg monotherapy during the Screening Phase.

Treatment Extension Phase begins once viral load from Treatment Visit 48 under PRO 140\_CD 03 study is available for Investigator review. The first Treatment Extension Visit (TE1) will take





place within 10 days of last treatment visit under CD03 study (i.e. T48 visit), with weekly visits  $(\pm 3 \text{ days})$  thereafter.

Study participants will be regularly monitored for viral load and will cease weekly study treatment injections should they experience virologic failure. Virologic failure is defined as two consecutive HIV-1 RNA levels  $\geq 200$  copies/mL.

All subjects who experience virologic failure at any time during the Treatment Extension Phase will undergo the Virologic Failure (VF) Visit assessments and then exit the Treatment Extension Phase to enter the Follow-up Phase of the study unless subjects receiving PRO 140 350mg or PRO 140 525mg opt to receive the higher dose of PRO 140 525mg or 700mg, respectively, for the remainder of Treatment Extension Phase. Subjects who do not experience virologic failure will complete EOT assessments and then enter the Follow-up Phase of the study at the end of Treatment Extension Phase.

Duration of Follow-up Phase is determined based on whether or not subject has experienced virologic failure during the Treatment Extension Phase.

Subjects receiving PRO 140 350mg who do not switch to PRO 140 525mg or subjects receiving PRO 140 525mg who do not switch to PRO 140 700mg, and all subjects receiving PRO 140 700mg who experience virologic failure during the Treatment Extension Phase will be assessed every 4 weeks until the viral suppression is achieved (i.e., plasma HIV-1 RNA levels decline to < 50 copies/mL). Additionally, virologic failure subjects will return to clinic for long-term follow-up at 6 months and at one year from the time of the Virologic Failure (VF) Visit.

Subjects who do not experience virologic failure at the end of Treatment Extension Phase, will be assessed every 2 weeks for a total of 4 weeks.

#### STUDY CENTER(S) 3.1

Site(s) participating in the PRO140 CD03 protocol

#### 3.2 STUDY POPULATION

Study population consists of virally suppressed HIV-1 patients with CCR5-tropic virus who complete the PRO140 CD03 study.

#### 3.3 **ELIGIBILITY CRITERIA**

### 3.3.1 Inclusion Criteria

Subjects must meet all of the following criteria to be included in the study:

- 1. Subjects who have completed 48 weeks of treatment in PRO140 CD03 study.
- 2. Last known Plasma HIV-1 RNA < 50 copies/mL within the PRO140 CD03 study.





- 3. Both male and female subjects and their partners of childbearing potential must agree to use 2 medically accepted methods of contraception (e.g., barrier contraceptives [male condom, female condom, or diaphragm with a spermicidal gel], hormonal contraceptives [implants, injectables, combination oral contraceptives, transdermal patches, or contraceptive rings], and intrauterine devices) during the course of the study (excluding women who are not of childbearing potential and men who have been sterilized). Females of childbearing potential must have a negative serum pregnancy test at Screening visit and negative urine pregnancy test prior to receiving the first dose of study drug.
- 4. Willing and able to participate in all aspects of the study, including use of SC medication, completion of subjective evaluations, attendance at scheduled clinic visits, and compliance with all protocol requirements as evidenced by providing written informed consent.

### 3.3.2 Exclusion Criteria

Potential subjects meeting any of the following criteria will be excluded from enrollment:

- 1. Not currently enrolled in PRO140\_CD03 study.
- 2. Any active infection or malignancy requiring acute therapy (with the exception of local cutaneous Kaposi's sarcoma).
- 3. Females who are pregnant, lactating, or breastfeeding, or who plan to become pregnant during the study.
- 4. Subjects weighing < 35kg.
- 5. History of anaphylaxis to any oral or parenteral drugs.
- 6. History of Bleeding Disorder or subjects on anti-coagulant therapy (except aspirin).

  Note: Subjects with well-controlled bleeding disorder while on stable anti-coagulant therapy dose with documented stable INRs can be enrolled as per discretion of the Investigator.
- 7. Any other clinical condition that, in the Investigator's judgment, would potentially compromise study compliance or the ability to evaluate safety/efficacy.





Figure 3-1: Study Flow Diagram





#### STUDY SCHEDULE

The study is divided into three phases: Screening, Treatment and Follow-up.

- 1. Screening Phase begins with signing of Informed Consent and lasts up to 21 days. Subject will enter the Treatment Extension Phase as soon as HIV-1 viral load and CD4 count results from T48 visit are available for review by Investigator.
- 2. Treatment Extension Phase begins with evaluation of results of laboratory samples collected during Screening Phase within the PRO140 CD03 study. The first treatment extension visit (TE1) will be administered within 10 days of treatment visit 48, with weekly visits ( $\pm$  3 days) thereafter.

All subjects will continue taking PRO 140 350mg, 525mg, or 700mg SC monotherapy during the Screening Phase.

Study participants will be regularly monitored for viral load during Treatment Extension phase, and will cease weekly study treatment injections should they experience virologic failure.

Subjects who experience virologic failure at any point during the Treatment Extension Phase will undergo the Virologic Failure (VF) Visit assessments and then exit the Treatment Phase to enter the Follow-up Phase of the study unless: subjects receiving PRO 140 350mg opt to receive PRO 140 525mg SC weekly injections and subjects receiving PRO 140 525mg opt to receive PRO 140 700mg SC for the remainder of Treatment Extension Phase.

Subjects who do not experience virologic failure will enter the Follow-up Phase of the study at the end of the Treatment Extension Phase.

- 3. Follow-Up Phase: The duration of follow-up depends on the status of viral load suppression.
  - Subjects receiving PRO 140 350mg or 525mg who do not elect to receive the higher dose of PRO 140 525mg or 700mg, respectively, in the Treatment Extension Phase and all subjects receiving PRO 140 700mg who experience virologic failure will be followed up every 4 weeks until viral suppression is achieved (i.e., plasma HIV-1 RNA levels to return to < 50 copies/mL). Additionally, virologic failure subjects will return to clinic at 6 months and at one year from the time of the Virologic Failure (VF) Visit.
  - Subjects who do not experience virologic failure at the end of Treatment Extension Phase. will be followed up every 2 weeks for a total of 4 weeks.

Procedures to be performed during each of these study phases are described below and provided as a Schedule of Assessments in Table 4-1 and Table 4-2.





Table 4-1: Schedule of Assessments – Screening and Treatment Extension Phase

| Procedure/Assessments | | Treatment Extension Phase | | | | In case of<br>Virologic Failure |
|---|---|---|---|---|---|---|
| | Screening | TE1 | | Subsequent | 9 | |
| Visit | Phase<br>(T46/47/48) | (Pre-Rx) | (Post-Rx) | TE Visits | EOT | VF |
| Window Period | Up to 21 days | Within 10 | days of T48 | Weekly ±3 days<br>from last treatment | | |
| Informed Consent <sup>[1]</sup> | X | | | - | ×. | |
| Physical Examination | $\mathbf{X}^{[2]}$ | X <sup>[3]</sup> | | X <sup>[3]</sup> | X | X |
| Neurological Assessment <sup>[4]</sup> | X | 115 | | 97 | X | Х |
| Vital Signs <sup>[5]</sup> | X | | X | X | X | X |
| ECG | X | 7: | | - | X | X |
| Complete Blood Count (CBC) <sup>[6]</sup> | X | | | X <sup>[19]</sup> | X | х |
| Biochemistry <sup>[7]</sup> | X | | | X <sup>[19]</sup> | X | х |
| Coagulation Indices | | | | X <sup>[19]</sup> | X | X |
| Urinalysis | | P | | X <sup>[19]</sup> | X | X |
| Urine Pregnancy Test <sup>[8]</sup> | | X | | | <br> | |
| Plasma HIV-1 RNA level <sup>[9]</sup> | X | X | | X | X | Х |
| TruCount T assay <sup>[9]</sup> | X | X | | Х | X | Х |
| Trofile® DNA Assay/PhenoSense® Entry | X | | | | X | X <sup>[10]</sup> |
| Trofile® RNA Assay/PhenoSense® Entry | | | | 80 | 38 | X <sup>[10]</sup> |
| PK sample for PRO 140 | X | | | X <sup>[11]</sup> | X | X |
| Anti-idiotypic Antibodies to PRO 140 | X | 1 | 1 | X <sup>[11]</sup> | X | X |
| HIV-1 Single Copy RNA Assay[12] | | X | | X <sup>[11]</sup> | X | |
| Genosure Archive Assay <sup>[13]</sup> | X | | | | X | Х |
| PhenoSense GT Assay <sup>[14]</sup> | | 20 | | × | DV | X |
| PRO 140 Administration <sup>[1]</sup> - 350mg SC - 525mg SC - 700 mg SC | X | | x | х | X | |
| Combination ART Regimen | | | | X <sup>[16]</sup> | X <sup>[16]</sup> | х |
| Injection Site Reaction Assessment <sup>[17]</sup> | | | X | Х | X | X |
| Adverse Events <sup>[18]</sup> | X | X | X | X | X | X |
| Concomitant Medications | X | X | X | X | X | X |
| CCR5 Receptor Occupancy <sup>[20]</sup> | | | | X | 58 | |




### X – Indicate assessments performed at T46/47/48 under PRO140 CD03 study

#### **Foot Notes:**

- (1) Informed consent must be obtained prior to patient participation in any protocol-related activities that are not part of routine care.
- (2) Complete physical performed by Investigator at SV, EOT or VF.
- (3) Symptom-directed physical examination performed at clinic visits.
- (4) The neurological assessment tool is based on the three question survey used by Simioni et al. (Simioni S, 2010). Additional neurological assessment modalities may be used as per Investigator's discretion.
- (5) Post-treatment vital signs (blood pressure, heart rate, respiration rate, and temperature) will be measured within 15 minutes of study treatment administration when visit performed at clinic.
- (6) Hemoglobin, Hematocrit (HCT), Red Blood Cells (RBC), White Blood Cells (WBC) with total and differential count, Absolute Neutrophil Count (ANC) and platelets.
- (7) Serum Biochemistry
  - o Hepatic function indicators: total and direct bilirubin, alkaline phosphatase, aspartate aminotransferase (AST), alanine aminotransferase (ALT), total protein, Lactate dehydrogenase (LDH)
  - o Renal function indicators: BUN, creatinine
  - o Electrolytes: sodium, potassium, chloride, calcium and bicarbonate
  - o Other: glucose (random), cholesterol (total)
- (8) ONLY performed on women of childbearing potential.
- (9) Plasma HIV-1 RNA and TruCount T Assay will be performed once every four (4) weeks when subject comes to clinic. TruCount T Assay includes: Absolute Lymphocytes, CD3 cell count, CD4 cell count, CD8 cell count, CD3%, CD4% and CD8%
- (10) Monogram Biosciences Trofile<sup>®</sup> DNA or RNA assay (or both) will be performed at the Virologic Failure Visit depending on the last known HIV-1 RNA levels, along with PhenoSense® Entry assay using AMD3100 (X4 inhibitor drug), Maraviroc and PRO 140 (R5 inhibitor drugs)
- (11) Sample will be collected at least once every eight (8) weeks when subject comes to clinic.
- (12) Single copy HIV-1 RNA Assay will be performed only if preceding viral load result is <20 copies/ml.
- (13) Monogram Biosciences GenoSure Archive Assay will be collected at SV, EOT, and in case of VF if last known HIV-1 RNA level is < 1000 copies/mL.
- (14) PhenoSense® GT (and PhenoSense Integrase and GeneSeq Integrase testing, if applicable, will also be collected if part of baseline ART regimen in PRO140 CD03 study) will be collected at VF visit if last known HIV-1 RNA level is >1000 copies/mL.
- (15) PRO 140 injections should be administered by qualified healthcare professional or self-administered by trained subjects
- (16) Baseline ART regimen will be restarted one week prior to final PRO 140 treatment visit and overlap with study treatment given at EOT or reinitiated at the time of virologic failure.
- (17) Injection Site Reaction Assessment as assessed by Investigator (or designee) at clinic visits and by visiting nurse or qualified medical professional during home visits. Injection Site Reaction Assessment will not be applicable if PRO 140 is self-administered by subjects at home.
- (18) Only AEs occurring after treatment injection at TE1 onwards will be captured, in addition to any ongoing AEs from PRO140 CD03 study.
- (19) To be collected every 12 weeks during the treatment extension phase.
- (20) Refer to Section 7.10.14.






# Table 4-2: Schedule of Assessments -Follow-Up (FU) Phase

# (a) Subjects who do NOT experience Virologic Failure

| Procedure/Assessments | Follow-Up Visit -1 | Follow-Up Visit -2 |
|---|---|---|
| | NVF-FU1 | NVF-FU2 |
| Window Period | 2 weeks<br>(±3 days) after EOT | 4 weeks<br>(±3 days) after EOT |
| Physical Examination | $X^{[1]}$ | $X^{[1]}$ |
| Vital Signs | X | X |
| Plasma HIV-1 RNA level | X | X |
| TruCount T assay | X | X |
| Anti-idiotypic Antibodies to PRO 140 | | X |
| Re-initiate combination Antiretroviral<br>Therapy | X | X |
| Adverse Events | X | X |
| Concomitant Medications | X | X |

<sup>[1]</sup> Symptom-directed physical examination

# (b) Subjects who experience Virologic Failure

# Short-Term Follow-Up Visits

| Procedure/Assessments | Follow-Up Visit -1 | Follow-Up Visit -2 | Follow-Up Visit -3 <sup>[1]</sup> |
|---|---|---|---|
| | VF-FU1 | VF-FU2 | VF-FU3 |
| Window Period | 4 weeks<br>(±7 days) after VF<br>visit | 8 weeks<br>(±7 days) after VF<br>visit | 12 weeks<br>(±7 days) after VF<br>visit |
| Physical Examination | $X^{[2]}$ | $X^{[2]}$ | $X^{[2]}$ |
| Vital Signs | X | X | X |
| Plasma HIV-1 RNA level | X | X | X |
| TruCount T assay | X | X | X |
| Anti-idiotypic Antibodies to PRO 140 | X | | |
| Re-initiate combination Antiretroviral<br>Therapy | X | X | X |
| Adverse Events | X | X | X |
| Concomitant Medications | X | X | X |

<sup>[1]</sup> Subject will be followed up every 4 weeks until viral suppression is achieved (i.e., plasma HIV-1 RNA levels decline to < 50 copies/mL). Subject will undergo additional follow-up visits every 4 weeks beyond VF-FU3 visit (up to a maximum of 6 months after re-initiation of combination antiviral therapy), if viral suppression is not achieved at the end of VF-FU3 visit.

# Long-Term Follow-Up Visits


<sup>[2]</sup> Symptom-directed physical examination

Version 5.0 Date: 30-Mar-2021



| Procedure/Assessments | Long-Term Follow-Up<br>Visit -1 | Long-Term Follow-Up<br>Visit -2 |
|---|---|---|
| | VF-6mFU | VF-12mFU |
| Window Period | 6 months (±1 month)<br>after VF visit | 12 months (±1 month)<br>after VF visit |
| Adverse Events <sup>[1]</sup> | X | X |
| Assessment of cART changes[2] | X | X |
| Plasma HIV-1 RNA level | X | X |
| TruCount T assay | X | X |
| Trofile® DNA or RNA Assay <sup>[3]</sup> | X | X |
| PhenoSense® Entry Assay <sup>[4]</sup> | X | X |
| HIV-1 Drug Resistance Assay <sup>[5]</sup> | X | X |

- Only SAEs and any AE that is considered possibly or probably or definitely related to the IP by the investigator will be captured during the long term follow up phase.
- [2] Any changes to the combination antiretroviral regimen since the viral re-suppression is achieved.
- [3] Monogram Biosciences Trofile® DNA or RNA (or both) assay will be performed depending on last known HIV-1 RNA levels.
- [4] Monogram Biosciences HIV-1 PhenoSense® Entry assay with AMD3100 (X4 inhibitor drug), Maraviroc and PRO 140 (R5 inhibitor drugs).
- [5] Monogram Biosciences GenoSure Archive Assay or PhenoSense® GT (and PhenoSense Integrase and GeneSeq Integrase testing, if applicable), will be performed depending on last known HIV-RNA levels.




#### 4.1 SCREENING PHASE

# 4.1.1 Screening Phase

The subject will sign and date the informed consent form (ICF) and Health Insurance Portability Accountability Act (HIPAA) authorization (according to site policy and practices) prior to any study-related procedures. The unique identification number (screening number) assigned under PRO140\_CD03 study will be retained.

All study centers will be instructed to maintain the study-specific screening and enrollment logs at their sites.

Once the ICF has been signed, screening procedures and information will be obtained to confirm subject eligibility including:

- Demographic information (see Section 7.3),
- Current medications review (see Section 7.5),
- Physical examination (see Section 7.6),
- Electrocardiogram (ECG) (see Section 7.7),
- Post-treatment vital signs (see Section 7.9),
- Collection of Blood Specimens (see Section 7.10) for
  - o Complete Blood Count
  - Biochemistry
  - o Plasma HIV-1 RNA level
  - TruCount T Assay
  - o PK sample for PRO 140
  - Anti-idiotypic Antibody for PRO 140
  - HIV-1 Drug Resistance Assay (GenoSure Archive<sup>®</sup> Assay)
  - o HIV-1 Co-Receptor Tropism (Trofile® DNA Assay)
    - CCR5 Genotyping will be tested using residual whole blood sample from tropism sample collected at Screening
  - o HIV-1 PhenoSense® Entry (Monogram BioSciences)

All screening information will be fully documented in the subject's medical records (i.e., source documents).




- For consented subjects who do not meet eligibility criteria, a Screen Failure electronic Case Report Form (eCRF) will be completed. The Screen Failure eCRF will contain the following details: the subject identification number, the date of ICF signature, demographic information (see Section 7.3), and the reason for screen failure. No additional information will be required for subjects who fail screening.
- For consented subjects who meet eligibility criteria, all required screening information will be transcribed onto the appropriate page of the eCRF.

Eligible subjects that are not enrolled within 21 days of Screening Visit will have Safety lab assessments repeated to reconfirm eligibility, with the exception of HIV-1 drug resistance, viral tropism and PhenoSense® Entry.

Note: Subjects who intend and consent to participate in Treatment Extension phase Study will not initiate ART Regimen therapy at T47.

#### 4.2 TREATMENT EXTENSION PHASE

Treatment Extension Phase begins with an evaluation of results of laboratory samples collected during the Screening Phase. Subjects who meet all eligibility criteria, as per data gathered from Screening Phase are to be treated. All subjects who fail to meet eligibility criteria will be considered screen failure and exit the study without further evaluation.

All subjects will continue receiving weekly dosing of PRO 140 350mg, 525mg, or 700mg monotherapy in the Treatment Extension Phase, given once per week (± 3 days), until virologic failure or another reason for discontinuation occurs, such as consent withdrawal or study drug approval, whichever occurs first. The study treatment (PRO 140 SC injections) will be administered by a qualified medical professional (MD, DO, PA, LPN, LVN, NP, RN, or CMA if state law permits) at clinic site, home visit, or self-administered by subjects. Study participants will be regularly monitored for viral load following initiation of PRO 140, and will cease weekly study treatment injections should they experience virologic failure.

As shown in Table 4-3, eligible subjects will be enrolled in one of the three treatment groups for treatment extension phase.

Table 4-3: Three Groups, Treatment Extension Phase

| Study Drug | Dosage<br>Form | IP<br>concentration | Dosing Frequency and Amount | Route of Administration |
|---|---|---|---|---|
| PRO 140<br>350mg | Parenteral solution | 175 mg/mL | 2 injections of PRO 140 (2 X 1 mL/inj.) | SC injection |
| PRO 140<br>525mg | Parenteral solution | 175 mg/mL | 2 injections of PRO 140 (2 X 1.5 mL/inj.) | SC injection |
| PRO 140<br>700mg | Parenteral solution | 175 mg/mL | 2 injections of PRO 140 (2 X 2 mL/inj.) | SC injection |






As shown in Figure 3-1, subjects receiving PRO 140 350mg or 525mg experiencing virologic failure in Treatment Extension Phase will have option of reinitiating ART regimen or beginning PRO 140 525mg or 700mg SC weekly injections, respectively, for the remainder of Treatment Extension Phase.

All subjects who experience virologic failure at any point during the Treatment Extension Phase will undergo the Virologic Failure (VF) Visit assessments and will be followed up every 4 weeks until viral suppression is achieved (i.e., plasma HIV-1 RNA levels decline to < 50 copies/mL). Virologic failure subjects will also return to clinic for long-term follow-up at 6 months and at one year from the time of the Virologic Failure (VF) Visit. Subjects who do not experience virologic failure will be followed up every 2 weeks for total of 4 weeks.

Study subjects will resume prior or alternate HAART regimen:

- One week prior to the end of Treatment Extension Phase, or
- Anytime during the Treatment Extension Phase, if virologic failure occurs or have met any other criteria for discontinuation of study treatment as specified in Section 5.2.1 of the protocol. Subjects will be allowed to continue PRO 140 monotherapy while waiting for new ART regimen to be constructed by the Investigator.

#### Note:

- Subjects may return to clinic for an additional blood draw in-between the clinic visits for plasma HIV-1 RNA levels, per the discretion of the Investigator.
- $\triangleright$  Virologic failure is defined as two consecutive levels of  $\ge 200$  copies/mL. Subjects experiencing virologic failure while on 350 mg or 525mg dose have option of re-initiating ART regimen or continuing the treatment with higher dose of PRO 140 (525mg SC or 700mg) weekly injection for remainder of Treatment Phase or until subsequent virologic failure event after viral re-suppression on higher dose. Subjects who meet any criteria (other than virologic failure) for discontinuation of study treatment as specified in Section 5.2.1 of the protocol, will undergo EOT Visit assessments and enter the Follow-up Phase of the study.
- > Subjects who do not experience virologic failure will enter the Follow-up Phase of the study at the end of Treatment Extension Phase.

Visits during the Treatment Extension Phase will commence on TE1, i.e. the date of first treatment, with weekly visits (± 3 days) thereafter. The first Treatment Extension Visit (TE1) will take place within 10 days of last treatment visit under CD03 study (i.e. T48 visit).




Note: Although the screening visit for CD03-Extn can be done at T46, 47, or 48 visit for CD03 study, all subjects must complete T48 treatment dosing under the CD03 study, before receiving first Treatment (at TE1 visit) under the CD03 Extension study.

# 4.2.1 Treatment Extension Phase: Treatment Extension Visit-1 (TE1)

The following assessments will be performed at TE1 visit, unless otherwise specified:

# **Pre-Treatment**

- Confirmation of eligibility criteria by reviewing test results and other criteria assessments performed at Screening Visit (see Section 7.2)
- Symptom-directed physical examination (see Section 7.6)
- Change in concomitant medications (see Section 7.5)
- Assessment of Adverse Events (AE) (see Section 9)
- Vital signs, pre- and post-treatment (see Section 7.9)
- Collection of blood specimens (see Section 7.10) for
  - o Plasma HIV-1 RNA level
  - TruCount T Assay
  - CCR5 Receptor Occupancy (IncellDx Lab)
  - HIV Drug Resistance Assay
  - o Plasma HIV-1 RNA Single Copy Assay
  - o PK sample for PRO 140
  - o Anti-idiotypic Antibody for PRO 140
- Urine pregnancy test (see Section 7.10.3)

### **Administration of PRO 140**

Study treatment will be administered as a subcutaneous injection in the abdomen.

Subjects will receive PRO 140 350mg, delivered as two 1 mL injections on opposite sides of the abdomen. PRO 140 525mg is delivered as two 1.5mL injections on opposite sides of the abdomen and PRO 140 700mg is delivered as two 2 mL injections on opposite sides of the abdomen.

Alternatively, the 525mg dose can be delivered as three 1mL injections (one injection on one side of the abdomen and two injections on the opposite side of the abdomen) or a single 3.0mL injection on either side of the abdomen, and the 700mg dose can be delivered as four 1mL injections (two injections on opposite sides of the abdomen)




**Note:** All treatment injections <u>must</u> be administered by a qualified medical professional (MD, DO, PA, LPN, LVN, NP, RN, or CMA if permitted by state law) at clinic site or home visit or self-administered by subjects, for the duration of the Treatment Extension Phase.

### **Post-Treatment**

- Injection Site Reaction Assessment (see Section 7.12)
  - Note: To assess injection site reactions, the Investigator will use the DAIDS AE grading table (refer to Section 16.3).
- Vital signs (see Section 7.9) will be assessed again within 15 minutes of study treatment administration.

# 4.2.2 Treatment Extension Phase: Subsequent Treatment Extension Visits

The following assessments will be performed at each treatment visit, unless otherwise specified:

- Assess for any Adverse Events and changes in Concomitant Medications (see Section 9 and 7.5),
- Symptom-directed physical examination (see Section 7.6),
- Vital Signs (see Section 7.9)
  - ➤ Note: Post-treatment vital signs will be assessed within 15 minutes following study treatment administration
- Collection of blood specimens (see Section 7.10) for
  - o Plasma HIV-1 RNA level
  - TruCount T Assay
    - ➤ **Note:** Blood sample for plasma HIV-1 RNA level and, TruCount T Assay should be collected at least once every four weeks starting from TE1 when subject comes to clinic.
  - Plasma HIV-1 RNA Single Copy Assay
  - o PK for PRO 140
  - Anti-idiotypic antibody for PRO 140
    - ➤ Note: Blood sample for plasma HIV-1 RNA Single Copy Assay, PK sample for PRO 140 and Anti-idiotypic antibody to PRO 140 should be collected at least once every eight weeks starting from TE1 when subject comes to clinic.
  - Complete Blood Count




- o Biochemistry
- Coagulation Indices
  - ➤ **Note:** Complete Blood Count, Biochemistry, and Coagulation Indices should be collected once every 12 weeks when subject comes to clinic.
- CCR5 Receptor Occupancy
  - Note: Blood will be taken prior to PRO 140 injection (trough sample) and 24-48 hours (peak sample) after the PRO 140 injection to check for CCR5 occupancy, and correlative analysis will be performed with PRO 140 PK concentration and HIV-1 RNA levels. This assessment will be performed up to 5 times at different treatment visits.
- Urinalysis
  - ➤ **Note:** Urinalysis should be collected once every 12 weeks when subject comes to clinic.
- Study treatment administration (PRO 140)
  - **Note:** All treatment injections <u>must</u> be administered by a qualified medical professional (MD, DO, PA, LPN, LVN, NP, RN, or CMA if permitted by state law) at clinic site or home visit or self-administered by subjects during the Treatment Extension Phase.
- Injection site reaction assessment (see Section 7.12)
  - ➤ **Note:** To assess injection site reactions, the Investigator will use the DAIDS AE grading table (refer to Section 16.3).
- Re-initiate previous antiretroviral regimen or an alternative regimen selected by the treating physician one week prior to EOT, if viral load remain suppressed.

# 4.2.3 Treatment Extension Phase: End of Treatment Visit (EOT)

The following assessments will be performed at End of Treatment (EOT) visit:

- Assess for any Adverse Events and changes in Concomitant Medications (see Section 9 and 7.5),
- Complete physical examination (see Section 7.6),
- Neurological assessment (see Section 7.8)
- Vital signs (see Section 7.9)
- Electrocardiogram (ECG) (see Section 7.7)




- Collection of blood specimens (see Section 7.10) for
  - o Complete Blood Count
  - o Biochemistry
  - Coagulation Indices
  - o Plasma HIV-1 RNA level
  - TruCount T Assay
  - o HIV-1 Single Copy RNA Assay
  - o HIV-1 Drug Resistance Assay (GenoSure Archive)
  - o Trofile DNA/RNA Assay
  - o PhenoSense® Entry Assay
  - o PK for PRO 140
  - Anti-idiotypic antibody for PRO 140
  - CCR5 Receptor Occupancy
- Urinalysis
- Study treatment administration (PRO 140)

**Note:** All treatment injections <u>must</u> be administered by a qualified medical professional (MD, DO, PA, LPN, LVN, NP, or RN) at clinic site or home visit or self-administered by subjects during the Treatment Extension Phase.

- Injection site reaction assessment (see Section 7.12)
  - ➤ **Note:** To assess injection site reactions, the Investigator will use the DAIDS AE grading table (refer to Section 16.3).
- Continue previous antiretroviral regimen or alternative regimen that was initiated <u>one week prior to EOT</u>, if viral load remain suppressed.

# 4.3 VIROLOGIC FAILURE (VF) VISIT

Virologic failure is defined as two consecutive levels of  $\geq 200$  copies/mL.

Subjects receiving PRO 140 350mg or 525mg that experience virologic failure have the option of re-initiating ART regimen or receiving a higher dose of PRO 140.

Subjects receiving 350 mg can increase their dose to 525mg for the remainder of the Treatment Extension Phase and those receiving 525 mg can increase their dose to 700 mg for the remainder




of the Treatment Extension Phase

The following assessments will be performed for subjects who experience virologic failure at any time during the Treatment Extension Phase prior to entering Follow-up Phase:

- Assess for any Adverse Events and changes in Concomitant Medications (see Section 9 and 7.5),
- Complete physical examination (see Section 7.6),
- Vital signs (see Section 7.9),
- Neurological assessment (see Section 7.8),
- Electrocardiogram (ECG) (see Section 7.7)
- Collection of blood specimens (see Section 7.10) for
  - Complete Blood Count
  - Biochemistry
  - o Plasma HIV-1 RNA level
  - TruCount T Assay
  - o HIV Drug Resistance Assay (PhenoSense GT)
  - o HIV Trofile® RNA/DNA Assay
  - o CCR5 Receptor Occupancy (IncellDx Lab)
  - o PhenoSense® Entry Assay
  - Quest Diagnostics Tropism Assay
  - o PK for PRO 140
  - Anti-idiotypic antibody for PRO 140
- Re-initiate previous antiretroviral regimen or an alternative regimen selected by the treating physician

# 4.4 FOLLOW-UP PHASE

The duration of follow-up depends on whether subject experiences virologic failure.

• Subjects who experience virologic failure within the Treatment Extension Phase will be assessed every 4 weeks until viral suppression is achieved (i.e., plasma HIV-1 RNA levels decline to < 50 copies/mL). Additionally, virologic failure subjects will return to clinic for




long-term follow-up at 6 months and at one year from the time of the Virologic Failure (VF) Visit

• Subjects who do not experience virologic failure at the end of the Treatment Extension Phase, will be assessed every 2 weeks for total of 4 weeks.

# 4.4.1 Follow-Up Visits

# 4.4.1.1 Short-Term Follow-Up Visits

# 4.4.1.1.1 Virologic Failure Subjects

Subjects who experience virologic failure during the Treatment Extension Phase will be assessed every 4 weeks until the viral suppression is achieved (i.e., plasma HIV-1 RNA levels decline to < 50 copies/mL).

The following assessments will be performed at each follow-up visit (VF-FU1, VF-FU2, VF-FU3 etc.), unless otherwise specified:

- Assess for any Adverse Events and changes in Concomitant Medications (see Section 9 and 7.5),
- Symptom-directed physical examination (see Section 7.6),
- Vital signs (see Section 7.9),
- Collection of blood specimens (see Section 7.10) for
  - o Plasma HIV-1 RNA level
  - TruCount T Assay
  - o Anti-idiotypic antibody for PRO 140 (VF-FU2 only)
- Continue previous antiretroviral regimen or an alternative regimen selected by treating physician

### 4.4.1.1.2 Non Virologic Failure Subjects

Subjects who do not experience virologic failure at the end of the Treatment Extension Phase, will be assessed every 2 weeks for total of 4 weeks.

The following assessments will be performed at each follow-up visit (NVF-FU1 and NVF-FU2 visits), unless otherwise specified:

- Assess for any Adverse Events and changes in Concomitant Medications (see Section 9 and 7.5),
- Symptom-directed physical examination (see Section 7.6),




- Vital signs (see Section 7.9),
- Collection of blood specimens (see Section 7.10) for
  - o Plasma HIV-1 RNA level
  - o TruCount T Assay
  - o Anti-idiotypic antibody for PRO 140 (NVF-FU2 only)
- Continue previous antiretroviral regimen or an alternative regimen selected by treating physician

# 4.4.1.2 Long-Term Follow-Up Visits

Additionally, subjects who experience virologic failure will also return to clinic for the long-term follow-up at 6 months and at one year from the time of the Virologic Failure Visit.

The following assessments will be performed at VF-6mFU and VF-12mFU visit, unless otherwise specified:

- Assess for any Adverse Events and changes in combination antiretroviral therapy (see Section 9 and 7.5)
  - Note: Only SAEs and any AE that is considered possibly or probably or definitely related to the study treatment by the Investigator will be captured during the long-term follow-up phase.
- Collection of blood specimens (see Section 7.10) for
  - o Plasma HIV-1 RNA level
  - TruCount T Assay
  - o HIV Drug Resistance Assay (PhenoSense GT)
  - o HIV Trofile® DNA or RNA Assay
  - o HIV PhenoSense Entry® Assay




# 5 SUBJECT COMPLETION AND WITHDRAWAL

### **5.1** SUBJECT COMPLETION

- A subject who completes the Treatment Extension Phase and 4-week Non-Virologic Failure Follow-Up Phase will be considered as having completed the study.
- A subject who experiences virologic failure during the Treatment Extension Phase, undergoes the Virologic Failure (VF) Visit assessments and is followed up until viral suppression is achieved in addition to completing the Virologic Failure 12 month Follow-Up (VF-12mFU) Visit, will be considered as having completed the study.

#### 5.2 SUBJECT WITHDRAWAL

A subject who enters the Treatment Extension Phase but does not complete the study, as defined in Section 5.1, is considered to have prematurely withdrawn from the Study.

All subjects have the right to withdraw at any point during treatment without prejudice to future care. It will be documented whether or not each subject completed the clinical study. If for any subject, study treatment or observations were discontinued, the reason(s) will be recorded.

The Investigator can discontinue a subject at any time if it is considered medically necessary.

In addition, subjects <u>WILL</u> be withdrawn from the study, in consultation with the Medical Monitor and the Investigator, if any of the following are met:

- A subject is significantly non-compliant with the requirements of the protocol
- The Investigator determines that it is in the best interest of the subject
- Subject chooses to withdraw or is withdrawn due to an adverse event
- Recurring Grade 2 study drug injection related AE at two consecutive visits
- Occurrence of Grade 3 study drug injection related AE
- A subject becomes pregnant

**Note**: The pregnancy will be followed to term for safety follow-up. Relevant safety information collected after the study has completed will be reported as supplemental information.

Discontinuation of study by Sponsor

Premature withdrawal from the study <u>MAY</u> occur if, in consultation with the Medical Monitor and the Investigator, any of the following are met:

- A subject is treated with a prohibited medication.
- Major protocol violation




### 5.2.1 Discontinuation of Study Treatment

Discontinuation of study treatment (PRO 140) and resumption of previous or alternative antiretroviral regimen is recommended if:

Subject experiences virologic failure (defined as two consecutive HIV-1 RNA levels of ≥ 200 copies/mL)

**Note**: Subjects receiving PRO 140 350mg or 525mg that experience virologic failure have the option of re-initiating ART regimen or receiving a higher dose of PRO 140 525mg or 700mg, respectively, for the remainder of the Treatment Extension Phase or until subsequent virologic failure event after viral re-suppression on higher dose.

- Develops AIDS-defining conditions as specified in Appendix I (Section 16.1) under which subject is unable to continue treatment with study drug (PRO 140), or subject require treatment with prohibited concomitant medications
- Shows signs or symptoms of clinically significant immunosuppression
- Subject or the subject's clinician wishes to restart ART
- Subject becomes pregnant

# 5.2.2 Data Collected for Withdrawn Subjects

Subjects may withdraw from the study or discontinue study treatment at any time; however, CytoDyn is dedicated to minimizing missing data in this study. It is therefore suggested that all subjects, regardless of whether they continue to receive study treatment, continue within the study.

Investigators considering discontinuing study treatment should contact the medical monitor prior to such discontinuation. Subjects who have study treatment discontinued will continue to be followed, per protocol, whenever possible. Subjects who have study treatment discontinued due to a serious adverse event will be followed until resolution or stabilization of the event.

In the event that a subject is withdrawn from the study at any time due to an adverse event or serious adverse event (SAE), the procedures stated in Section 9.1.1 or 9.2.1, respectively must be followed.

Every attempt should be made to collect follow-up information. The reason for withdrawal from the study will be recorded in the source documents and on the appropriate page of the eCRF.

Before a subject is identified as lost-to-follow up, the site should make all reasonable efforts to contact the subject. These attempts must be documented and should include at a minimum one phone call and one certified letter.

#### 5.3 SCREEN FAILURES






A subject who has signed a consent form, but is not treated is classified as a screen failure. Subject number, demographics and reason for screen failure will be recorded.

If a subject initially fails to meet inclusion/exclusion criteria and is later reconsidered for participation, the subject will be re-consented and retain the unique screening number assigned under the PRO 140 CD 03 study.




#### 6 STUDY TREATMENT

#### 6.1 INVESTIGATIONAL PRODUCT DESCRIPTION

PRO 140 is a humanized IgG4, k monoclonal antibody (mAb) to the chemokine receptor CCR5. PRO 140 is provided at a concentration of 175 mg/mL and is intended for SC route of administration.

Kits will be labeled with a unique identification number. Each kit used during the Treatment Phase will contain vials of PRO 140 for SC injection. For the 350 mg dose, one milliliter (1 mL) of PRO 140 solution will be drawn from each vial and loaded into the syringe. A total of 350mg, 525mg, or 700mg (175 mg/mL) of PRO 140 is delivered as two 1 mL, 1.5 mL, or 2mL injections, respectively, administered subcutaneously on opposite sides of the abdomen or as one of the alternative methods listed in the table below. One study injection kit will be assigned per subject per treatment, except for 350mg dose in which one kit can be used for 2 visits. Each vial of the PRO 140 product contains ~1.4 or 2.4 mL antibody at 175mg/mL in a buffer containing 5 mM L-histidine, 15.0 mM glycine, 95 mM sodium chloride, 0.3% (w/v) sorbitol, 0.005% (w/v) polysorbate 20 (Tween 20®), and sterile water for injection, at pH of 5.5.

| PRO 140 Kits Containing 1.4 mL per Vial | | | | |
|---|---|---|---|---|
| PRO 140<br>Dose | # of Vials<br>Used per<br>Dose | Total Injection Volume (mL) | Volume (mL) Administered per Injection* | Volume (mL) Discarded per Vial |
| 350 mg | 2 | 2 | 1 | 0.4 |
| 525 mg | 3 | 3 | 1.5 | 0.4 |
| 700 mg | 4 | 4 | 2 | 0.4 |
| PRO 140 Kits Containing 2.4 mL per Vial | | | | |
| PRO 140<br>Dose | # of Vials<br>Used per<br>Dose | Total Injection Volume (mL) | Volume (mL) Administered per Injection* | Volume (mL) Discarded per Vial |
| 350 mg | 1** | 2 | 1 | 0.4 |
| 525 mg | 2 | 3 | 1.5 | 0.9 |
| 700 mg | 2 | 4 | 2 | 0.4 |




<sup>\*</sup>When 2 injections given per dose; 1 injection on opposite sides of the abdomen.

**Note:** For the 350 mg dose, 1 mL injection will be drawn from 1.4 mL solution in a vial. Remaining 0.4 mL medication will be discarded appropriately from each vial. For the 525 mg dose, 1 mL will be drawn from 1.4 mL solution in vial #1, and 0.5 mL will be drawn from 1.4 solution in vial #2 for a total of 1.5 mL injection per side. For the 700 mg dose, 1 mL will be drawn from 1.4 mL solution from vial #1, and 1 mL will be drawn from 1.4 mL solution in vial #2 for a total of 2 mL injection per side.

Alternatively, when 2.4 mL vials are provided, 1.5 or 2 mL injection will be drawn and the remaining will be discarded from each vial. Subjects in both group B and C will require two vials for a single dose. Unused content of PRO 140 in a vial should remain in the vial and **not** be administered to any other subject.

Table 6-1 provides the unit strength, dosing frequency and mode of administration for the study drug.

| Study Drug | Dosage<br>Form | IP<br>concentration | Dosing Frequency and Amount | Route of<br>Administration |
|---|---|---|---|---|
| PRO 140<br>350mg | Parenteral solution | 175 mg/mL | 2 injections of PRO 140 (2 X 1 mL/inj.)<br>per week on opposite sides of abdomen<br>during Treatment Extension Phase | SC injection |
| PRO 140<br>525mg | Parenteral solution | 175 mg/mL | 2 injections of PRO 140 (1.5 mL/inj.)<br>per week on opposite sides of abdomen<br>during Treatment Extension Phase | SC injection |
| PRO 140<br>700mg | Parenteral solution | 175 mg/mL | 2 injections of PRO 140 (2 mL/inj.)<br>per week on opposite sides of abdomen<br>during Treatment Extension Phase | SC injection |

Table 6-1: Investigational Product - PRO 140

# 6.2 INVESTIGATIONAL PRODUCT PACKAGING AND LABELING

Study drug will be prepared by Ajinomoto Althea, Inc. and will be packaged, labeled, and shipped by PCI Clinical Services.

The contents of each vial are described in Section 6.1. PRO 140 kits will be labeled with information such as: study protocol #; fill volume; concentration; storage condition; a "use as per study protocol" statement; a cautionary statement; sponsor's name and address; and the kit number.

Below are representative samples of the Investigational Product, FDP individual vial (Figure 6-1), syringe label (Figure 6-2), and kit labels (


<sup>\*\*</sup>Since each vial contains 2.4 mL of PRO 140 only 1 vial is needed for the 350 mg dose. The second vial can be utilized to administer 350 mg dose at the subsequent visit.





Figure 6-3) designated for use in this clinical protocol. Each 350mg kit contains two labeled vials and syringe labels, and each 525mg kit contains three labeled vials and syringe labels. The 700mg dose will consist of two 350mg kits (4 labeled vials and syringes total).

Figure 6-1: PRO 140 (CHO) 175mg/mL - Vial Label

| Protocol: PRO 140_CD03/Ext Kit N | No. xxxxx | Protocol: PRO 140_CD03/Ext | Kit No. xxxxx |
|---|---|---|---|
| Subject No | | Subject No. | |
| Single use 3 mL vial contains 1.4 mL of PRO mg/mL) solution for subcutaneous injection | 140 (175 | Single use 3 mL vial contains 1.4 mL of mg/mL) solution for subcutaneous inject | |
| Store at 2°C to 8°C (36°F to 46°F) | | Store at 2°C to 8°C (36°F to 46°F) | |
| USE AS PER STUDY PROTOCOL | | USE AS PER STUDY PROTOCOL | |
| Caution: New Drug – Limited by Federal (or U<br>Law to Investigational Use | Jnited States) | Caution: New Drug – Limited by Federa<br>Law to Investigational Use | 1 (or United States) |
| CytoDyn Inc., Vancouver, WA, USA | | CytoDyn Inc., Vancouver, WA, USA | |
| Protocol: PRO 140_CD03/Ext Kit N | No. xxx | Protocol: PRO 140_CD03/Ext | Kit No. xxx |
| Subject No | | Subject No. | |
| Single use 3 mL vial contains 2.4 mL of PRO mg/mL) solution for subcutaneous injection | 140 (175 | Single use 3 mL vial contains 2.4 mL of mg/mL) solution for subcutaneous inject | , |
| Store at 2°C to 8°C (36°F to 46°F) | | Store at 2°C to 8°C (36°F to 46°F) | |
| USE AS PER STUDY PROTOCOL | | USE AS PER STUDY PROTOCOL | |
| Caution: New Drug – Limited by Federal (or U<br>Law to Investigational Use | Jnited States) | Caution: New Drug – Limited by Federa<br>Law to Investigational Use | 1 (or United States) |
| CytoDyn Inc., Vancouver, WA, USA | | CytoDyn Inc., Vancouver, WA, USA | |

Figure 6-2: PRO 140 (CHO) 175mg/mL - Syringe Label

Protocol: PRO 140\_CD03/Ext

Contents of Kit No. xxxxx

This syringe contains 1mL, 1.5mL, or 2mL PRO 140 (175 mg/mL) solution for subcutaneous injection

USE AS PER STUDY PROTOCOL

Caution: New Drug – Limited by Federal (or United States) Law to Investigational Use

CytoDyn Inc., Vancouver, WA, USA




Protocol: PRO 140 CD03/Ext

Contents of Kit No. xxxxx

Kit No. xxxxx

This syringe contains 1.5 mL PRO 140 (175 mg/mL) solution for subcutaneous injection

USE AS PER STUDY PROTOCOL

Caution: New Drug – Limited by Federal (or United States) Law to Investigational Use

CytoDyn Inc., Vancouver, WA, USA

Protocol: PRO 140 CD03/Ext

Figure 6-3: PRO 140 (CHO) 175mg/mL - Kit Label

| Site No | Subject No. |
|---|---|
| This kit contains 2 single-use vials | |
| Each 3 mL vial contains 1.4 mL of PRO 140 (175 mg/mL) solution for subcutaneous injection | |
| Store at 2°C to 8°C (36°F to 46°F) | |
| USE AS PER STUDY PROTOCOL | |
| Caution: New Drug – Limited by Federal (or United States) Law to Investigational Use | |
| CytoDyn Inc., Vancouver, WA, USA | |
| Protocol: PRO 140_CD03/Ext | Kit No. xxxxx |
| Site No | Subject No. |
| This kit contains 3 single-use vials | |
| Each 3 mL vial contains 1.4 mL of PRO 140 (175 mg/mL) solution for subcutaneous injection | |
| Store at 2°C to 8°C (36°F to 46°F) | |




#### USE AS PER STUDY PROTOCOL

Caution: New Drug – Limited by Federal (or United States) Law to Investigational

Use

CytoDyn Inc., Vancouver, WA, USA

| Protocol: PRO 140_CD03 | Kit No. xxx |
|---|---|
| Site No | Subject No. |
| This kit contains 2 single-use vials | |
| Each 3 mL vial contains 2.4 mL of PR subcutaneous injection | O 140 (175 mg/mL) solution for |
| Store at 2°C to 8°C (36°F to 46°F) | |
| USE AS PER STUDY PROTOCOL | |
| Caution: New Drug – Limited by Fede Use | eral (or United States) Law to Investigational |
| CytoDyn Inc., Vancouver, WA, USA | |

NOTE: Subjects with low body fat percentages may find subcutaneous injections uncomfortable esp. in case of 1.5 mL or 2 mL injection for the 525mg or 700mg dosing. In such cases, PRO 140 525 mg can be injected as three 175mg/ml injections and PRO 140 700mg can be injected as four 175mg/ml injections and/or subcutaneous injections can be placed at different areas other than abdomen as per discretion of the Investigator.

The pharmacy manual provides the criteria regarding vial acceptance or rejection, as well as instructions for the preparation of the IP syringes to be used to administer drug.

#### 6.3 INVESTIGATIONAL PRODUCT STORAGE

Study drug will be shipped at 2°C to 8°C (refrigerated [36°F to 46°F]) to the Investigator's site. Upon receipt at the site, the responsible site staff or pharmacist should verify the integrity of the vials. Study drug should be stored at 2°C to 8°C (refrigerated [36°F to 46°F]). The contents of the vial should appear as a clear to opalescent, colorless to yellow solution; fine translucent particles may be present. This is normal.

The Investigator must maintain an accurate record of the shipment, storage, and dispensing of the study drug in a drug accountability log. An accurate record including the date and amount of study drug dispensed for each subject must be available for inspection at any time. A study CRA assigned






to monitor the investigational site will review these documents once study drug has been received by the investigational site. Study drug will be accounted for on an ongoing basis during the study.

#### 6.4 INVESTIGATIONAL PRODUCT ADMINISTRATION

Guidelines for dose preparation can be found in the pharmacy manual.

PRO 140 will be provided to the administering personnel in single-use syringes prepared from vials of study drug stored at 2-8°C at the site pharmacy prior to use. Each of two syringes is filled to deliver 1 mL, 1.5 mL, or 2 mL of study drug.

Equivalent volumes of study drug will be administered subcutaneously on opposite sides of the abdomen. However, based on subject preference or investigator discretion subjects receiving each of the doses can be administered using an alternate approach as follows:

# 350mg Dose:

• One 2 mL injection on one side of the abdomen.

# 525mg Dose:

- One 3 mL injection on one side of the abdomen.
- Three 1 mL injections, two on one side of the abdomen and one on the other side.

### **700 mg Dose:**

• Four 1 mL injections, on opposite sides of the abdomen, or other location.

A 25-guage needle should be used to remove IP from vial and for administration to subjects, and drug should not be held in syringe for longer than 1 hour.

IP should be administered slowly over 15 seconds per mL.

Following each SC delivery of drug, careful examination will be made to assess the appearance of any study drug Injection Site Reactions (ISRs) as described in Section 16.3.

All doses of study drug will be administered as SC injection by a qualified medical professional (MD, DO, PA, LPN, LVN, NP, RN, or CMA if state law permits) at clinic site or home visit or self-administered by subjects.

**Note:** It is preferred that the same area of the abdomen be used throughout the study. At the same time, it is not recommended to inject the study drug into areas where skin shows signs of a previous injection site reaction. It is advised to change the injection site if any previous injection site reaction remains unresolved

#### 6.5 INVESTIGATIONAL PRODUCT RECEIPT AND ACCOUNTABILITY






Study drug must be used in accordance with this protocol and only under the direction of the responsible Investigator. The investigational site must maintain complete and accurate records showing receipt and disposition of all study drug, including master records listing the date of receipt, the number and nature of medication units received, and a dispensing record which includes each quantity dispensed, identification of the staff member/subject to whom dispensed, the date of dispensing, the intended study participant, and the identification of the preparer. All used and unused study kits will be retained by the investigational site until drug accountability can be confirmed by study CRA during the monitoring visits. Instructions will be provided by Sponsor regarding final disposition of all study drug in compliance with applicable regulations.

#### 6.6 INVESTIGATIONAL PRODUCT DISPOSITION

All drug supplies are to be used only for this protocol and not for any other purpose. The Investigator must not destroy any drug labels or any partially used or unused drug supply until instructed by the Sponsor. At the conclusion of the study and as appropriate during the course of the study, the Investigator will return all used and unused drug containers and drug labels to the drug distributor as directed by the Sponsor. A copy of the completed drug disposition form will be sent to CytoDyn, Inc. or to its designee.




#### 7 DESCRIPTION OF PROTOCOL ASSESSMENTS AND PROCEDURES

### 7.1 INFORMED CONSENT

Written informed consent will be obtained for this study by the Investigator or designee from all subjects before the performance of any protocol-specific procedure. This study will be conducted in accordance with the provisions of the Declaration of Helsinki.

In obtaining and documenting informed consent, the Investigator must comply with applicable regulatory requirements and must adhere to Good Clinical Practice (GCP). The Investigator, or designee, must fully inform subjects of all pertinent aspects of the study. Before informed consent may be obtained, the Investigator, or a person designated by the Investigator, must provide the subject ample time and opportunity to inquire about details of the study and to decide whether or not to participate in the trial. All questions about the trial must be answered to the satisfaction of the subject. Prior to the subject's participation in the trial, the written informed consent must be signed and personally dated by the subject and by the person who conducted the informed consent discussion. Authorization for release of protected health information must also be obtained, as per local policies.

#### 7.2 ASSESSMENT OF ELIGIBILITY

During the Screening Visit and at TE1 Visit (prior to treatment administration), the Investigator must assess a subject's continued suitability and eligibility for the trial. The Inclusion and Exclusion criteria of this Protocol are described in Sections 3.3.1 and 3.3.2. If the subject is not suitable or eligible for the trial then the subject will be a screen failure.

### 7.2.1 Re-screening

If a subject initially fails to meet inclusion/exclusion criteria, and is later reconsidered for participation, the subject will be re-consented and retain the unique screening number assigned under PRO 140\_CD 03 study.

#### 7.3 DEMOGRAPHIC INFORMATION

For the purposes of this study, demographic information will include:

- Dates of ICF signature
- Date of birth
- Gender
- Race (American Indian/Alaskan Native, Asian, Black/African American, Native Hawaiian/Pacific Islander, Caucasian, or other)




• Ethnicity (Hispanic/Latino or Not Hispanic/Latino)

#### 7.4 MEDICAL HISTORY

Medical history will be brought forward from PRO140\_CD03 study.

#### 7.5 CONCOMITANT MEDICATIONS AND NON-STUDY TREATMENTS

Prior medications/therapies will be brought forward from PRO140 CD03 study.

Subjects must be questioned at each study visit concerning any new medications or changes in current medications including over-the-counter medication.

For each medication and non-study treatment, the following will be documented:

- Medication/treatment name (generic name may be used if trade name is unknown)
- Dose, unit, and frequency of dosing (individual dosages, not total daily dose).
  - Note: Each new dose of medication should be recorded as a separate entry, with the exception of medications that are given on a sliding scale. For these, it is acceptable to enter the range of the dosage, including the start and stop dates for which the specified dosage range was used.
- Route of dosing
- Indication for use
- The start date
- The stop date (if medication/therapy is not ongoing)

Please refer to Exclusion Criteria (Section 3.3.2) for a list of prohibited treatments and/or procedures. All other medications that are appropriate for the care of the subject may be prescribed. If concomitant medications are started during the study, the indication for the concomitant medication should be considered an AE.

# 7.5.1 Excluded Medications and Therapies

1. Use of concomitant antiretroviral therapy is NOT allowed during the Treatment Extension Phase of the study EXCEPT for one week overlap of existing retroviral regimen and PRO 140 at the end of the treatment in subjects who do not experience virologic failure. Subject is allowed to re-initiate antiretroviral therapy during the Treatment Extension Phase, if virologic failure occurs or if subject meets any other criteria for discontinuation of study treatment as specified in Section 5.2.1 of the protocol.




- 2. Use of oral or parenteral corticosteroids (> 5 mg/day) is NOT allowed during the study, with the following exceptions:
  - Use of chronic systemic corticosteroids at replacement doses (e.g., < 5mg/day prednisone) AND use of inhaled, nasal, or topical steroids are allowed.
  - Use of short course of systemic corticosteroids (Medrol pack) after TE2 will only be allowed with prior approval from the sponsor.
- 3. Use of radiation or cytotoxic chemotherapy, immunosuppressants and immunomodulating agents (e.g., interleukins, interferons) or agents with known anti-HIV activity (i.e., hydroxyurea, foscarnet) are NOT allowed during the study.
- 4. Use of any non-FDA approved/investigational therapy

# 7.5.2 Allowable Medications and Therapies

All other medications/therapies that are not otherwise prohibited and, in the judgment of the Investigator, are required for proper medical care of the subject may be prescribed.

#### 7.6 PHYSICAL EXAMINATION

The complete physical examination will include routine examinations for the following:

- General Appearance
- Head, Ears, Eyes, Nose, Throat (HEENT)
- Lymph Nodes
- Heart/Cardiovascular abnormalities
- Respiratory
- Abdomen
- Genitourinary
- Musculoskeletal and Extremities
- Neurologic abnormalities
- Dermatologic abnormalities
- Any other body system for which an abnormality is noted and which, in the opinion of the Investigator, is relevant to the safety of the subject or could impact safety or efficacy results for the subject; i.e., the abnormality is clinically significant (CS).

Each abnormality will be recorded and the Investigator will record an assessment of its clinical significance.




The complete physical examination will be conducted at the Screening Visit (SV), End of Treatment Visit (EOT) and at Virologic Failure (VF) Visit. Only symptom-directed physical examination will be performed at scheduled and unscheduled treatment and follow-up visits conducted within the clinic.

# 7.7 ELECTROCARDIOGRAM

A resting 12-lead ECG will be conducted at the Screening Visit (SV) and at EOT/VF visit and the results will be evaluated by the Investigator. Only those subjects who have normal or not-clinically significant results at the Screening Visit (SV) will be enrolled in this study.

The following parameters will be recorded: ventricular rate (beats per minute), PR interval (msec), QRS interval (msec), QT interval (msec), and QTc interval (msec). Additionally, the Investigator will record the overall results of the ECG reading as either normal or abnormal, and as either not clinically significant or clinically significant. If abnormalities are observed, each will be recorded.

#### 7.8 NEUROLOGICAL ASSESSMENT

Neurological assessment will be performed by the Principal Investigator or Study Coordinator at SV and EOT/VF Visit.

The neurological assessment tool is based on the three question survey used by Simioni et al. [Simioni S, 2010]. Refer to Section 16.4 for further details. Additional neurological assessment modalities may be used as per Investigator's discretion.

#### 7.9 VITAL SIGNS

Vital signs will be collected at all study visits performed at the clinic. Vital signs collected during the Treatment Extension Phase will be performed post-treatment, and assessed within 15 minutes following study treatment administration.

The following vital signs will be collected at all visits, unless otherwise stated:

- Seated blood pressure (taken after the subject has been seated for at least 5 minutes)
- Heart Rate
- Respiration Rate
- Temperature

# 7.10 CLINICAL LABORATORY ASSESSMENTS

Blood and urine samples will be collected according to the time points in the schedule of assessments for analysis of the following parameters:




#### 7.10.1 Routine CBC

- <u>Frequency of testing</u>: At SV, at least once every twelve (12) weeks during Treatment Extension Phase, EOT or VF
- Includes hemoglobin, hematocrit (HCT), red blood cell (RBC) count, white blood cell (WBC) count, WBC differential count (%), absolute neutrophils count and platelets count.

# 7.10.2 Biochemistry

- <u>Frequency of testing</u>: At SV, at least once every twelve (12) weeks during Treatment Extension Phase, EOT or VF
- Biochemistry profile includes assessment of:

<u>Hepatic function indicators:</u> total and direct bilirubin, alkaline phosphatase, aspartate aminotransferase (AST), alanine aminotransferase (ALT), total protein, LDH

Renal function indicators: BUN, creatinine

Electrolytes: sodium, potassium, chloride, calcium and bicarbonate

Other: glucose (random), cholesterol (total)

# 7.10.3 Coagulation Indices

- <u>Frequency of testing</u>: At least once every twelve (12) weeks during Treatment Extension Phase, EOT, or VF
- Prothrombin time (PT) and International Normalized Ratio (INR)

# 7.10.4 Urinalysis

- <u>Frequency of testing</u>: At least once every twelve (12) weeks during Treatment Extension Phase, EOT, or VF
- Urine samples will be tested for color, appearance, specific gravity, pH, protein, glucose, occult blood, ketones, leukocyte esterase, nitrite, bilirubin, urobilinogen, and microscopic examination of urine sediment

# 7.10.5 Urine pregnancy test

- Frequency of testing: At TE1 prior to first treatment administration
- A urine sample will be collected from female subjects of childbearing potential. This test will be performed at the study site using a commercially available kit.

# 7.10.6 Plasma HIV-1 RNA level and TruCount T Assay




- <u>Frequency of testing</u>: At SV, prior to administration of PRO 140 at Treatment Extension Visit 1 (TE1), at least once every four (4) weeks during Treatment Extension Phase, EOT, and at VF visit when subject comes to clinic. In addition, blood sample will also be collected at all Virologic Failure Follow-up (VF-FU) and Non-Virologic Failure Follow-up (NVF-FU) visits.
- To assess antiretroviral therapeutic response to PRO 140 or cART regimen

**Note:** Plasma HIV-1 RNA level will be measured using Human Immunodeficiency Virus 1 (HIV-1), Quantitative, RNA (Taqman® Real-Time PCR) test.

TruCount T Assay includes measurement of Absolute Lymphocytes, CD3 cell count, CD4 cell count, CD8 cell count, CD3%, CD4% and CD8%

# 7.10.7 HIV-1 Trofile® DNA Assay

- Frequency of testing: At SV, EOT/VF visits, in addition to VF-6mFU and VF-12mFU visits if last known HIV-1 RNA level is <1000 copies/mL.
- To assess HIV-1 co-receptor tropism. This test determines eligibility for CCR5 antagonist therapy for patients infected with HIV-1. Only those subjects who have exclusive CCR5-tropic virus will be eligible to participate in this study.
- Unlike the standard Trofile® assay (which uses viral RNA), Trofile® DNA Assay can determine the coreceptor tropism of a patient's HIV-1 strain when the patient's viral load is undetectable.

# 7.10.8 HIV-1 Trofile® RNA Assay

• Frequency of testing: At VF, VF-6mFU and VF12mFU Visits, if last known HIV-1 RNA level is >1000 copies/mL.

#### 7.10.9 HIV-1 Drug Resistance Assay

- a. GenoSure Archive Assay
  - o GenoSure Archive assay provides HIV-1 antiretroviral drug resistance data when standard resistance testing cannot be performed due to inadequate plasma viral load.
  - o <u>Frequency of sample collection</u>: At SV, and, EOT at VF, VF-6mFU and VF-12mFU visits, if last known HIV-1 RNA level is <1000 copies/mL.

# b. PhenoSense® GT

PhenoSense® GT is a combination resistance test for three classes of antiretroviral drugs (i.e., nucleoside/nucleotide, non-nucleoside, and protease inhibitors), that provides both




phenotypic and genotypic results from the same blood sample (viral load  $\geq$ 500 copies/mL).

- o <u>Frequency of sample collection</u>: At VF, VF-6mFU and VF-12mFU visits, if last known HIV-1 RNA level is >1000 copies/mL.
- c. PhenoSense Integrase and GeneSeq Integrase testing

PhenoSense Integrase and GeneSeq Integrase testing will be additionally performed in conjunction with PhenoSense® GT, if subject has past exposure to an integrase or in cases where complex drug resistance patterns is known or suspected.

Samples for PhenoSense® GT (and PhenoSense Integrase and GeneSeq Integrase testing, if collected) will be stored at Lab and will be analyzed only if subject experiences virologic failure.

# 7.10.10 Plasma HIV-1 RNA Single Copy Assay

- <u>Frequency of sample collection</u>: At TE1 prior to first treatment administration and at least once every eight (8) weeks during Treatment Extension Phase, if last known viral load is < 20 copies/mL, and EOT.
- To assess antiretroviral therapeutic response to PRO 140 cART regimen

# 7.10.11 PK sample for PRO 140

• <u>Frequency of testing:</u> At SV, at least once every eight (8) weeks during Treatment Extension Phase, EOT/VF visits.

# 7.10.12 Anti-idiotypic antibodies to PRO 140

<u>Frequency of sample collection</u>: At SV, at least once every eight (8) weeks during Treatment Extension Phase, EOT/VF visits Additionally, sample will be collected at Virologic Failure Follow-up Visit 1 (VF-FU1) and Non-Virologic Failure Follow-up Visit 2 (NVF-FU2)

#### 7.10.13 PhenoSense® Entry Assay

- Frequency of testing: At SV, EOT, VF, VF-6mFU and VF-12mFU visits in conjunction with tropism assessment
- With AMD3100 (X4 inhibitor drug), Maraviroc and PRO 140 (R5 inhibitor drugs).

# 7.10.14 CCR5 Receptor Occupancy

• To assess the number CCR5 receptors on patients' CD4 cell surface. Of those CCR5 receptors, the test will also assess the number and percentage of CCR5 receptors that are covered by PRO 140.




• Frequency of testing: This assessment will be performed up to 5 times at different treatment visits. Blood will be taken prior to PRO 140 injection (trough sample) and 24-48 hours (peak sample) after the PRO 140 injection to check for CCR5 occupancy, and correlative analysis will be performed with PRO 140 PK concentration and HIV-1 RNA levels

# 7.10.15 All laboratory reports will be reviewed by the Investigator.

Post-treatment abnormal results that are considered by the Investigator to be clinically significant will be recorded as adverse events. If the Investigator judges it necessary, testing may be repeated in order to make the determination of clinical significance. Validated, quality-controlled laboratory data will be transferred to the main database for analyses.

#### 7.11 PRO 140 ADMINISTRATION

Refer to Section 6.4 for details.

#### 7.12 INJECTION SITE REACTION ASSESSMENT

At each treatment visit that occurs at the clinical site, an injection site reaction assessment will be made for the current and previous injection sites. Injection site reaction assessments are recorded by the Investigator starting after the first injection is given. Refer to Sections 9.1.8 and 16.3 for more details.

# 7.13 COVID-19 GUIDANCE

The purpose of this guidance is to inform sites how to proceed in light of the challenges faced by patients and clinical trial sites as a result of COVID-19 shelter-in-place mandates from state governments. The content of this letter is based on FDA Guidance on Conduct of Clinical Trials of Medical Products during COVID-19 Pandemic (18 Mar 2020).

- The current schedule of assessments requires subjects to visit the clinic at least once every four weeks for lab assessments. Subjects may still continue to receive treatment with PRO 140 if they are unable to visit the clinic.
- Site staff may visit subjects' homes to conduct study assessments and/or deliver PRO 140.
- Sites may ship PRO 140 to subjects' homes if subjects are unable to visit the clinic.
- If subjects are unable to visit the clinic at least once every four weeks lab assessments will be missed. If this occurs site staff should contact subjects weekly by phone to assess:
  - Compliance to study treatment
  - Potential adverse events
  - Changes in concomitant medications






- Sites should document phone calls and include confirmation of compliance to study treatment, and report any adverse events and/or changes in medications.
- Subjects who report positive tests results for COVID-19 should have the diagnosis recorded as an adverse event.
- Sites should clearly document reasons for failing to obtain required assessments (e.g., limitation imposed by COVID-19 leading to the inability to perform the protocol-specified assessment).
- Any changes in the study visit schedule or missed visit should be entered as protocol
  deviation in the EDC and reason should be documented as missed study visit or visit
  performed out of window period due to COVID-19.
- If subject is early withdrawn from the study due to COVID-19, the reason should be clearly documented in the End of Study (EOS) section in EDC as "study discontinuation due to COVID-19".
- Monitoring activities will be performed remotely until Centers for Disease Control (CDC) recommendations allow travel to resume.




#### 8 STATISTICAL CONSIDERATIONS

This section presents general information about statistical considerations and concepts such as statistical power, sample size, and a brief discussion on analysis methodology, as well as some data conventions. Detailed descriptions of the statistical analysis methods and data conventions that will be used in this study will be in a separate document; i.e., the Statistical Analysis Plan (SAP).

#### 8.1 TREATMENT GROUPS

All eligible subjects in the study will receive PRO 140 as a 350mg, 525mg, or 700mg subcutaneous injection weekly.

#### 8.2 DESCRIPTION OF STUDY OUTCOME MEASURES

# **8.2.1** Primary Outcome Measures

The primary outcome measures for this study are:

- To assess the long term clinical safety of PRO 140 monotherapy regimen
- Proportion of participants experiencing virologic failure for all subjects and within each treatment group

# **8.2.2** Secondary Outcome Measures

There are multiple secondary outcome measures to be assessed in this study:

- Time to virologic failure for all subjects and within each treatment group
- Proportion of participants achieving viral re-suppression (HIV-1 RNA < 50 copies/mL) after experiencing virologic failure for all subjects and within each treatment group
- Time to achieving viral re-suppression (HIV-1 RNA < 50 copies/mL) after experiencing virologic failure for all subjects and within each treatment group
- Proportion of virologic failure subjects achieving viral re-suppression with re-initiation of previous baseline antiretroviral regimen for all subjects and within each treatment group
- Mean change in CD4 cell count, at each visit within the Treatment Phase for all subjects and within each treatment group

**Note:** Virologic failure is defined as two (2) consecutive plasma HIV-1 RNA levels of  $\geq 200$  copies/mL.

# 8.2.3 Safety Assessments

Safety measurements will include:

• Tolerability of repeated subcutaneous administration of PRO 140 as assessed by Investigatorevaluation of injection site reactions for all subjects and within each treatment group.




- Frequency of Grade 2, 3 or 4 adverse events as defined by the DAIDS Adverse Event scale
- Frequency of treatment–emergent serious adverse events

#### 8.3 SAMPLE SIZE DETERMINATION AND RATIONALE

Sample size determination is not applicable as only those subjects who are currently enrolled in PRO 140\_CD 03 study are allowed to participate in this study.

#### 8.4 RANDOMIZATION AND BLINDING

This study is an open label study with two treatment arms with no randomization and blinding requirements.

#### 8.5 Interim Analysis

No planned interim analysis.

#### 8.6 GENERAL STATISTICAL CONSIDERATIONS

# 8.6.1 Analysis Populations

The **Safety** population is defined as all subjects who received at least one dose of PRO 140. This population will be used for the analysis of primary and secondary outcome measures for this study.

#### **8.6.2** Statistical Methods

All collected study data will be presented in subject data listings. Statistical analyses will be performed using SAS® for Windows, version 9.4 or later.

A SAP will be developed and approved before the database is locked. The SAP will present the detailed statistical methodology to be used in analyzing the efficacy and safety data from this trial.

#### **8.6.3** Prognostic Factors/Covariates

Not applicable.

# 8.6.4 Handling of Missing Data

There will be no imputation of missing data for this study.

#### 8.6.5 Multicenter Study

This is a multicenter clinical trial.

#### 8.7 DATA SUMMARY

# 8.7.1 Subject Disposition






The disposition of all subjects who sign an ICF will be provided. The number of subjects screened, received treatment, completed, and discontinued during the study, as well as the reasons for all post treatment discontinuations will be summarized. Disposition and reason for study discontinuation will also be provided as a by-subject listing.

# 8.7.2 Demographic and Baseline Characteristics

Demographics and baseline characteristics (i.e., Age, Gender, Time since HIV diagnosis, Viral load at Screening Visit, etc.) will be summarized using appropriate descriptive statistics.

Medical history of the subjects will also be provided as a by-subject listing.

#### 8.7.3 Prior and Concomitant Medications

Prior and concomitant medications will be summarized for the Safety population. All prior and concomitant medications recorded in the eCRFs will be coded to generic term and all matching Anatomic Therapeutic Classification (ATC) codes using WHO Drug Summaries will be prepared using the coded terms. All prior and concomitant medications recorded in the eCRFs will also be listed.

# 8.7.4 Efficacy Analysis

All data from the primary and secondary outcome measures will be summarized and tabulated according to the variable type:

- Continuous data summaries will include number of observations, mean, standard deviation, median, and minimum and maximum values.
- Categorical data summaries will include frequency counts and percentages.

#### 8.7.5 Safety Analysis

The Safety population will be used for the analysis of safety assessments.

For continuous variables data will be summarized using n, mean, Standard Deviation (SD), minimum and maximum values. For categorical variables data will be summarized using frequency and percentage.

# 8.7.5.1 Adverse Events

Adverse events will be coded using Medical Dictionary for Regulatory Activities (MedDRA). TEAEs are defined as events with an onset on or after the first treatment. TEAEs will be summarized by treatment group, System Organ Class, and preferred term. The following TEAE summaries will be provided:

- TEAEs by severity grade
- TEAEs by relationship to study treatment.




In addition, separate summaries of SAEs, and AEs resulting in discontinuation of study treatment will be presented.

# 8.7.5.2 Tolerability Assessment

All data from tolerability assessments of repeated subcutaneous administration of PRO 140 as assessed by Investigator-evaluation of injection site reactions will be summarized.

# 8.7.5.3 Clinical Laboratory Data

All laboratory values will be listed. Laboratory measurements will also be summarized.

# 8.7.5.4 Physical Examination

All physical examination findings will be listed and any abnormality will be summarized.

# 8.7.5.5 Vital Signs

All vital sign assessment findings will be listed and summarized.

#### 8.7.5.6 ECG Examination

All ECG examination findings will be listed and any abnormality will be summarized.

# 8.7.5.7 Neurological Assessment

All neurological assessment findings will be listed and any abnormality will be summarized.






# ADVERSE EVENTS (DEFINITIONS AND REPORTING)

The Investigator is responsible for the detection and documentation of events meeting the criteria and definition of an AE or SAE, as provided in this protocol. During the study when there is a safety evaluation, the Investigator or site staff will be responsible for detecting, documenting, and reporting AEs and SAEs as detailed in this section of the protocol.

#### 9.1 ADVERSE EVENT

An adverse event (AE) is defined as any unfavorable or unintended sign, symptom, or disease that occurs or is reported by the subject to have occurred, or a worsening of a pre-existing condition. An AE may or may not be related to the study treatment.

AEs will be elicited through direct questioning and subject reports. Any abnormalities in visit evaluations, physical examination findings or laboratory results that the Investigator believes are clinically significant to the research subject and that occurred after initiation of the first study treatment will be reported as AEs. Abnormal findings that are NOT clinically significant (NCS) should not be recorded as an AE.

#### **Reporting of Adverse Events** 9.1.1

Report initiation for all AEs and SAEs will begin at the time of the first treatment extension visit and continue up until the final study visit (i.e. up to NVF-FU2 for subject who do not experience virologic failure or until viral suppression is achieved for subjects who experience virologic failure). Additionally, virologic failure subjects will have a long-term follow-up visits at 6 months and at one year from the time of the Virologic Failure Visit. Only SAEs and any AE that is considered possibly or probably or definitely related to the study treatment by the Investigator will be captured during the Long-term Follow-up Phase of the study. All events will be followed to resolution or until 30 days after the subject completes the study. A final assessment of outcome will be made at that time.

All AEs must be recorded in the subject's medical records and on the eCRFs. AEs will be reported using customary medical terminology along with the following information: the onset and end dates, whether the event is considered to be a SAE (see Section 9.2), the impact the event had on study treatment (see Section 9.1.2 ), the DAIDS AE grade (intensity) of the event (see Section 9.1.3), the causality of the event (see Section 9.1.4), whether treatment was given as a result of the event (see Section 9.1.5), and the outcome of the event (see Section 9.1.6).

#### 9.1.2 Impact of Study Treatment

The impact the event had on the study treatment will be assessed as either: none, study treatment interrupted, study treatment discontinued, or not applicable. The "not applicable" assessment will






be used only when the subject is no longer in the treatment phase of the protocol, or if the outcome of the event was "death".

# 9.1.3 DAIDS AE Grade (Severity) Assessment

The Investigator will carefully evaluate the comments of each subject and the response to treatment in order to judge the true nature and severity of the AE. The question of the relationship of AEs to study drug should be determined by the Investigator after thorough consideration of all available facts. To assess severity, the Investigator will use the DAIDS AE grading table (for adverse events as well as any injection site reactions refer to Section 16.2 and Section 16.3).

The general guidelines for assessing the AE grade appear below. Full guidelines may be obtained at

http://rsc.techres.com/Document/safetyandpharmacovigilance/DAIDS\_AE\_Grading\_Table\_v2\_N OV2014.pdf.

Grade 1 indicates a mild event

Grade 2 indicates a moderate event

Grade 3 indicates a severe event

Grade 4 indicates a potentially life-threatening event

Grade 5 Death related to AE.

Table 9-1: DAIDS AE Grading General Guidelines

DAIDS AE Grading Table Version 2.0- November 2014

#### 9.1.4 Causality Assessment

Adverse events will be assigned a relationship (causality) to the study treatment. The Principal Investigator (PI) must review each AE and make the determination of relationship of the event to the study treatment. Relationship of AEs to study treatment will be classified as follows:

- 1. Definitely related: This category applies to those AEs that the Investigator feels are incontrovertibly related to the study treatment. An AE may be assigned an attribution of definitely related if or when it meets all of the following criteria: (1) it follows a reasonable temporal sequence from administration of the study treatment; (2) it could not be reasonably explained by the known characteristics of the subject's clinical state, environmental or toxic factors, or other modes of therapy administered to the subject; (3) it follows a known response pattern to treatment with the study treatment.
- 2. Probably related: This category applies to those AEs which, after careful medical consideration at the time they are evaluated, are felt with a high degree of certainty to be






related to the study treatment. An AE may be considered probable if or when (must have three): (1) it follows a reasonable temporal sequence from administration of the study treatment. (2) It could not readily have been produced by subject's clinical state, environmental or toxic factors, or other therapies administered to the subject. (3) Disappears or is decreased upon discontinuation of the study treatment. (4) It follows a known response pattern to treatment with the study treatment.

- 3. **Possibly related**: This category applies to those AEs which, after careful medical consideration at the time they are evaluated, are judged unlikely but cannot be ruled out with certainty to the study treatment. An AE may be considered possible if or when (must have two): (1) it follows a reasonable temporal sequence from administration of the study treatment. (2) It could not readily have been produced by subject's clinical state, environmental or toxic factors, or other therapies administered to the subject. (3) Disappears or is decreased upon discontinuation of the study treatment. (4) It follows a known response pattern to treatment with the study treatment.
- 4. **Remotely related**: In general this category can be considered applicable to those AEs which, after careful medical consideration at the time they are evaluated, are judged likely to be unrelated to the study treatment. An AE may be considered unlikely if or when (must have two): (1) it does not follow a reasonable temporal sequence from administration of the study treatment. (2) It could not readily have been produced by subject's clinical state, environmental or toxic factors, or other therapies administered to the subject. (3) Disappears or is decreased upon discontinuation of the study treatment. (4) It does not follow a known response pattern to treatment with the study treatment.
- 5. **Unrelated**: This category applies to those AEs which, after careful consideration at the time they are evaluated, are clearly and incontrovertibly due to extraneous causes (disease, environment, etc.) and determined with certainty to have no relationship to the study treatment.

#### 9.1.5 Treatment Given as a Result of the Event

The event impact in terms of treatment provided will be as either: none, medication administered, non-medication therapy administered, surgery, or other (with a specification).

# 9.1.6 Outcome Assessment

The outcome of the event will be assessed as either: resolved, resolved with sequelae, ongoing, or death. Only one AE per subject is allowed to have an outcome assessment as "death." If there are multiple causes of death for a given subject, only the primary cause of death will have an outcome of death.




# 9.1.7 Expected / Anticipated Adverse Events

The most common potential study drug-related adverse reaction reported is mild headache. Other adverse events likely to be related to the drug include mild to moderate diarrhea, nausea, and fatigue.

# 9.1.8 SC Injection-related Events

SC and IV injections of concentrated protein materials can be associated with injection-related AEs that impact the ability to safely and successfully deliver the drug. Local injection-site reactions may include pain/discomfort, induration, erythema, nodules/cysts, pruritus, ecchymosis, etc. For SC injections, bleeding, absorption of the drug, leakage of drug, and induration at the local injection site can be additional complications. Other AEs that are common to monoclonal antibody-based therapies are chills, headache, backache, malaise, fever, pruritus, rash, nausea, tingling, and hypertension.

SC injection-related events will be monitored according to the guidelines provided in Section 16.2 (Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events [DAIDS AE Grading Table]). Injection-site reactions thought to be directly related to the injection are considered to be AEs of special interest, and a separate guideline for the acquisition of data related to this AE of special interest is provided in Section 16.3.

For subjects who develop grade 1 event or first occurrence of grade 2 events, continue therapy as per protocol. If a subject chooses to discontinue study treatment, the site should notify the protocol team leadership, and encourage the subject to complete any remaining study visits until the toxicity resolves.

For subjects who develop grade 2 event following study drug injection, the subject should be reevaluated closely until the AE returns to Grade ≤1, at which time study treatment may be reintroduced at the discretion of the site Investigator. If the same Grade 2 AE recurs following the next administration of study drug, study treatment must be permanently discontinued. Subjects experiencing Grade 3 AEs requiring permanent discontinuation of study treatment should be followed closely for resolution of the AE to Grade  $\leq 2$  and the team leadership must be notified.

Subjects with Grade 3 asymptomatic laboratory abnormalities in cholesterol, creatine kinase (CK) or triglycerides may continue study treatment.

For grade 4 events permanently discontinue therapy.

#### SERIOUS ADVERSE EVENTS (SAE) 9.2

A SAE is defined as any AE that:

Results in death




- Is life threatening (the subject is at immediate risk of dying from the AE)
- Requires subject hospitalization or prolongs existing hospitalization
- Results in persistent or significant disability/incapacity
- Is a congenital anomaly/birth defect

Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered a serious adverse event when, based upon appropriate medical judgment, they may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.

If a pregnancy occurs in a subject or partner of a male subject during the study, it must also be reported to CytoDyn, Inc. Any pregnant subject must be followed up by the Investigator or designee until the child is born. Any complication experienced through the end of the pregnancy should be considered as an adverse event (AE), and should be recorded, and if it meets the seriousness criteria, it must be reported to CytoDyn, Inc/designated CRO promptly. Participants who become pregnant will be entered into the Antiretroviral Pregnancy Registry (http://www.apregistry.com).

# 9.2.1 Reporting of Serious Adverse Events

The Investigator is required to report all SAEs that occur during the time period specified in Section 9.1.1. Once the Investigator becomes aware of an SAE, the SAE should be submitted to within 24 hours:



The may request additional supporting documentation as it becomes available, such as lab reports, ECG reports, discharge summary, hospital notes, etc.

The Investigator is also responsible for reporting all SAEs to the appropriate Institutional Review Board (IRB) in accordance with local laws and regulations. The Investigator is responsible for maintaining documentation in the study file that indicates the IRB has been properly notified. Under 21 CFR 312.32(c), the sponsor is required to notify FDA and all participating investigators in an IND safety report (i.e., 7- or 15-day expedited report) of potentially serious risks from clinical trials or any other source as soon as possible, but no later than 15 calendar days after the sponsor receives






the safety information and determines that the information qualifies for reporting. Participating investigators include all Investigators to whom the sponsor is providing drug under any of its INDs or under any investigator's IND (21 CFR 312.32(c)(1)).

# 9.2.2 SAE Follow-Up

All subjects experiencing an SAE, including the discontinued subjects, must be closely followed until sufficient information is obtained to indicate a return to normal status or until the event stabilizes at a level acceptable to the Investigator (i.e., recovery, return to baseline status, no further improvement expected, or death).

For each SAE indicated as an unresolved event on the initial report, regardless of whether the subject completed the study or withdrew, the site should submit a follow-up report with updated information.






#### 10 DIRECT ACCESS TO SOURCE DATA/DOCUMENTATION

Subjects will be identified on eCRFs by a unique subject identification number and on source documents by name/initials and date of birth. No personal identifier will be used in any publication or communication used to support this research study. The subject identification number will be used if it becomes necessary to identify data specific to a single subject.

The monitors, auditors, personnel authorized by the Sponsor, the local IRB, and the FDA are eligible to review medical and research records related to this study as a part of their responsibility to protect human subjects in clinical research and will be given direct access to source data and documentation (e.g., medical charts/records, printouts etc.) for source data verification, provided that subject confidentiality is maintained in accordance with local requirements. Access to electronic medical records may be governed by institution policy and each site will be required to ensure access while remaining compliant with institutional requirements.






#### 11 QUALITY CONTROL AND QUALITY ASSURANCE

#### 11.1 MONITORING REQUIREMENTS

In an effort to fulfill the obligations outlined in 21 Code of Federal Regulations (CFR) Part 312 and ICH guidelines which requires the Sponsor to maintain current personal knowledge of the progress of a study, the Sponsor's designated monitor will visit the center(s) during the study as well as maintain frequent telephone and written communication. The Investigator will permit the Sponsor to monitor the study as frequently as is deemed necessary and provide access to medical records to ensure that data are being recorded adequately, that data are verifiable and that protocol adherence is satisfactory.

The Investigator will permit representatives of the Sponsor and/or designated CRO to inspect all eCRFs and corresponding study subject original medical records (source documents) at regular intervals throughout the study. Subject original medical records and other relevant data must be available to support all data recorded in the eCRF. In addition to the original medical records, these data may include but are not limited to, study, laboratory and diagnostic reports, neurological assessment results, etc.

Site inspections serve to verify strict adherence to the protocol and the accuracy of the data being entered on the case report forms, in accordance with federal regulations. A Monitoring Log will be maintained at each study site which the monitor will sign, date and state the type of visit.

The Investigator should be aware that the study site and subject records may be inspected by the Sponsor and or representatives of the designated CRO, FDA or other regional regulatory authority.

For the IA, a cut-off date for data collection and monitoring will be determined and sites will be requested to provide current information up to the cut-off date.

# 11.2 ACCEPTABILITY OF CASE REPORT FORMS (CRFs)

Electronic CRFs must be completed for each subject who has signed an informed consent form. For subjects who are screen failures, this would be limited to the screen failure eCRF page. All source documents and eCRFs will be completed as soon as possible after the subject's visit. Corrections to data on the eCRFs will be documented. The Investigator will review eCRFs to indicate that, to his/her knowledge, they are complete and accurate. Electronic CRFs will be reviewed by the Sponsor's or designated CRO's monitor, who will make a decision as to their acceptability.

#### 11.3 MODIFICATION OF PROTOCOL

The Investigator will not modify or alter this protocol without first obtaining the concurrence of the Sponsor.






Approval by the Investigator's IRB must also be obtained prior to implementation of the change, with two exceptions:

- 1. When necessary to eliminate apparent immediate hazard to the subject; or
- 2. When the modification does not involve the subject's participation in the trial.

An amendment may also require modification of the informed consent form. The Investigator will provide an approval letter for the amendment and revised informed consent form, if applicable, to the Sponsor. An amendment must be in writing and it must be dated by both the Sponsor and the Investigator. If necessary, the Sponsor will submit protocol amendments to FDA and other appropriate regulatory authorities and notify other Investigators using this protocol.

#### 11.4 REPORTING PROTOCOL DEVIATIONS

The Investigator is obligated to follow the protocol without departure from the requirements written in the protocol. If the Investigator deviates from the protocol requirements, the Sponsor will make the determination as to whether the subject will continue in the study. The Sponsor also has the right to discontinue the subject for protocol violations. The IRB may also have to be contacted if safety to the subject or if the scientific soundness of the study is involved. All protocol deviations must be documented in the eCRFs.






# 12 ETHICS AND REGULATORY REQUIREMENTS

This study is to be conducted in accordance with the specifications of this protocol and in accordance with principles consistent with Declaration of Helsinki, GCP, 21 CFR Part 312, ICH E6, HIPAA regulations in 45 CFR Part 164 (US only), and the Belmont Principles of respect for persons, beneficence, and justice. No protocol changes will be implemented without the prior review and approval of the IRB, except when the modification does not involve the subject's participation in the trial or where it may be necessary to eliminate an immediate hazard to a research subject. In the latter case, the change will be reported to the IRB as soon as possible, according to IRB regulations.

Additionally, all study products used in this study are manufactured, handled and stored in accordance with applicable GMP and the products provided for this study will be used only in accordance with this protocol.

#### 12.1 Institutional Review Board/Independent Ethics Committee (IRB/IEC)

The Principal Investigator at the site will provide the Institutional Review Board/Independent Ethics Committee (IRB/IEC) with all appropriate materials as required by their IRB/IEC, including but not limited to the clinical study protocol, informed consent form, and any advertising materials. The study will not be initiated until the IRB/IEC provides written approval of the aforementioned documents and until approval documents have been obtained by the Principal Investigator and Sponsor or Sponsor designee. The Investigator will not participate in the decision. If the Investigator is an IRB or IEC member, documentation must be provided indicating recusal from the approval process. Appropriate reports on the progress of this study by the Principal Investigator will be made to the IRB/IEC as required by local and applicable government regulations and in agreement with policy established by the Sponsor. The Investigator is required to maintain an accurate and complete record of all written correspondence to and received from the IRB/IEC, and must agree to share all such documents and reports with the Sponsor.

No changes from the final approved protocol will be initiated without the IRB/IEC's prior written approval or favorable opinion of a written amendment, except when necessary to eliminate immediate hazards to the subjects or when the modification does not involve the subject's participation in the trial.

#### 12.2 Investigator's Responsibilities

The Investigators are responsible for performing the study in full accordance with the protocol and the current revision of the Declaration of Helsinki, the Good Clinical Practice: Consolidated Guideline, approved by the ICH, and any applicable national and local laws and regulations.






Information regarding any study centers participating in this study that cannot comply with these standards will be documented

#### 12.3 SUBJECT INFORMED CONSENT REQUIREMENTS

Written and oral information about the study in a language understandable by the subject will be given to all subjects by the Investigator and/or designee. Written informed consent will be obtained from each subject before any procedures or assessments that would not otherwise be required for the care of the subject are done and after the aims, methods, anticipated benefits, potential hazards, and insurance arrangements in force are explained and the subject has been given sufficient time to ask questions and consider participation in the study. It will also be explained to the subjects that they are free to refuse entry into the study and free to withdraw from the study at any time without prejudice to future treatment. It is permissible for a third person (e.g., a family member) to be present during the explanation of the study.

The written Informed Consent Form ICF is to be in compliance with CFR 21 Part 50.27 and GCP guidelines. The Sponsor and/or designated CRO will approve the ICF and all amendments to the ICF prior to submission to the IRB/IEC. A copy of the ICF to be used will be submitted by the Investigator to the IRB/IEC for review and approval prior to the start of the study. Each study site must provide the Sponsor with an unsigned copy of IRB/IEC-approved ICF along with applicable documentation to support this approval. The original signed ICF is retained in the subject's study records, and a copy is provided to the subject. A second copy may be filed in the subject's medical record, if allowed by institutional policy.




#### 13 DATA HANDLING AND RECORD KEEPING

#### 13.1 RECORDING AND COLLECTION OF DATA

The primary source document for this study will be the subject's medical record. If separate research records are maintained by the Investigator(s), the medical record and the research records will be considered the source documents for the purposes of auditing the study.

Applicable source data will be manually transcribed to the approved eCRFs. The Investigator is ultimately responsible for the accuracy of the data transcribed on the forms. All source documents and eCRFs will be completed as soon as possible after the subject's visit.

The Investigator will review eCRFs to indicate that, to his/her knowledge, they are complete and accurate. Designated source documents will be signed and dated by the appropriate study personnel. The Investigator must agree to complete and maintain source documents and eCRFs for each subject participating in the study.

All research data will be entered, either electronically or manually, into a computerized database. The clinical database will be designed by the clinical data manager in accordance with 21 CFR Part 11 and based on protocol requirements defined by the Sponsor in association with the Lead Investigator.

The Investigator will maintain a confidential list of study subjects that will include each subject's study number, name, date of birth, and unique hospital identification number if applicable. This list will be kept by the Investigator and will not be collected by the Sponsor. A notation will be made in the subject's case history/medical chart that he/she is participating in a clinical study and has provided a signed and dated ICF as well as a release for protected health information as required by local policies. The Investigator must also maintain a separate screening log of all the subjects screened for participation in the study; it should include gender, age, eligibility status, reason for ineligibility, if applicable; and study allocated subject number, if applicable.

# 13.2 CLINICAL DATA MANAGEMENT

The Sponsor and/or designated CRO will be responsible for the processing and quality control (QC) of the data. Data management will be carried out as described in the Sponsor's or CRO's standard operating procedures (SOPs) for clinical studies.

The handling of data, including data QC, will comply with regulatory guidelines (e.g., ICH E6 GCP, and local regulations where applicable) and the Sponsor's or the CRO's SOPs as well as provisions of the study-specific Data Management Plan.

#### 13.3 ARCHIVING






All study documentation at the Investigator site and Sponsor site will be archived in accordance with ICH GCP E6 and the Sponsor's quality standards and SOPs.

The Investigator will maintain all research records, reports, and case history reports for a period of two years after regulatory approval of the investigational product. If no application is filed or if the application is not approved, records must be maintained for two years after all investigations have been completed, terminated or discontinued and the FDA has been notified.

These documents should be retained for a longer period however, if required by the applicable regulatory requirements or if needed by Sponsor or its authorized representative (as per GCP 5.5.11).

At the completion of the study, details of the archival process must be provided to the Sponsor. Study records are subject to inspection by applicable health and regulatory agencies at any time.

Records to be retained by the Investigator include, but are not restricted to:

- Source data and the primary records upon which they are based (e.g., subject's progress notes, adverse event data, test results, and any other diagnostic procedures required to evaluate the progress of the study)
- Completed CRFs
- Signed protocols and protocol amendments
- Laboratory results, ranges, and certifications
- Product (e.g., IP supplies) and accountability records
- Study personnel signature log
- Monitoring logs
- Correspondence to and from the Sponsor, designee and IRB
- Investigator and Sub-Investigator CVs
- Signed informed consent and protected health information consent forms
- Subject screening and enrollment log
- SAE reports
- IRB approval and re-approval letters
- Other documents pertaining to the conduct of the study

These documents must be maintained and kept on file by the Investigator so that the conduct of the study can be fully documented and monitored.

At the completion of the study, details of the archival process must be provided to the Sponsor. Study records should not be transferred from site or destroyed without prior written agreement between the Sponsor and the study Investigator.






#### 14 PUBLICATION PLAN

All information supplied by CytoDyn in connection with this study and not previously published, is considered confidential information. This information includes, but is not limited to, the Investigator's Brochure (IB), clinical protocol, case report forms and other scientific data. Any data collected during the study are also considered confidential. This confidential information shall remain the sole property of CytoDyn, shall not be disclosed to others without the written consent of CytoDyn, and shall not be used except in the performance of this study.

It is understood by the Investigator that the Sponsor will use the information collected in this clinical trial in connection with the development of PRO 140. Therefore, this information may be disclosed as required to other Investigators or appropriate regulatory authorities. By agreeing to participate in this clinical trial, the Investigator understands that he/she has an obligation to provide the Sponsor with complete test results and all data developed during this trial.

**Publication and Disclosure**: Because this is a multi-center trial, the site and Investigator shall not independently publish, publicly disclose, present or discuss any results of or information pertaining to the site's and Investigator's activities conducted under this protocol until such multi-center publication is released with the written approval and under the direction of Sponsor. Notwithstanding the foregoing, if a multi-center publication is not released within eighteen (18) months after completion of analysis of all study data from all studies conducted within the multicenter trial, both the site and Investigator shall have the right to publish the results of and information pertaining to the site's and Investigator's activities conducted under this protocol and the clinical trial agreement, subject to the prior review and written approval of Sponsor. The site and Investigator agree to submit any proposed manuscript, presentation or other public disclosure regarding the study to Sponsor for review at least thirty (30) days prior to submitting such proposed manuscript to a publisher or delivering or making such presentation or other public disclosure to any third party. Within thirty (30) days of its receipt, Sponsor shall advise the site and/or Investigator, as the case may be, in writing of any information contained therein that is confidential information (other than research results included in a proposed manuscript) or that may impair Sponsor's ability to obtain patent protection. Sponsor shall have the right to require the site and/or Investigator, as applicable, to remove specifically identified confidential information (but may not require removal of research results from a proposed manuscript) and/or to delay the proposed submission or delivery of the proposed manuscript or presentation, or other public disclosure, for an additional sixty (60) days to enable Sponsor to seek patent protection. The site and Investigator shall not publish, publicly disclose, present or discuss any results of or information pertaining to the site's and Investigator's activities prior to completion of the trial, even if the multi-center trial or the study is terminated before its completion and the final clinical study report is signed off, or with respect to any outcome measures or analyses other than those specified in this protocol.






#### 15 REFERENCES

Arribas JR Pulido F, Delgado R, Lorenzo A, Miralles P, Arranz A, González-García JJ, Cepeda C, Hervás R, Paño JR, Gaya F, Carcas A, Montes ML, Costa JR, Peña JM. Lopinavir/ritonavir as single-drug therapy for maintenance of HIV-1 viral suppression: 48-week results of a randomized, controlled, open-label, proof-of-concept pilot clinical trial (OK Study). J Acquir Immune Defic Syndr.. - 2005. - Vol. 40. - pp. 280-287.

Boffito M Back DJ, Hoggard PG, Caci A, Bonora S, Raiteri R, Sinicco A, Reynolds HE, Khoo S, Di Perri G. Intra-individual variability in lopinavir plasma trough concentrations supports therapeutic drug monitoring. AIDS. - 2003. - Vol. 17. - pp. 1107-1108.

Cahn P Montaner J, Junod P, Patterson P, Krolewiecki A, Andrade-Villanueva J, Cassetti I, Sierra-Madero J, Casiró AD, Bortolozzi R, Lupo SH, Longo N, Rampakakis E, Ackad N, Sampalis JS. Pilot, randomized study assessing safety, tolerability and efficacy of simplified LPV/r maintenance therapy in HIV patients on the 1st PI-based regimen. PLoS One.. - 2011. - Vol. 6. - p. e23726.

**Calza L Manfredi R.** Protease inhibitor monotherapy as maintenance regimen in patients with HIV infection. Curr HIV Res.. - 2012. - Vol. 10. - pp. 661-72..

Cameron DW da Silva BA, Arribas JR, Myers RA, Bellos NC, Gilmore N, King MS, Bernstein BM, Brun SC, Hanna GJ. A 96-week comparison of lopinavir-ritonavir combination therapy followed by lopinavir-ritonavir monotherapy versus efavirenz combination therapy. Infect Dis.. - 2008. - Vol. 198. - pp. 234-240.

**Demeter LM Shafer RW, Meehan PM, Holden-Wiltse J, Fischl MA, Freimuth WW, Para MF, Reichman RC.** Delavirdine susceptibilities and associated reverse transcriptase mutations in human immunodeficiency virus type 1 isolates from patients in a phase I/II trial of delavirdine monotherapy (ACTG 260). Antimicrob.Agents Chemother.. - 2000. - Vol. 44. - pp. 794-797.

Guiguet M Ghosn J, Duvivier C, Meynard JL, Gras G, Partisani M, Teicher E, Mahamat A, Rodenbourg F, Launay O, Costagliola D and CO4. FHDH-ANRS Boosted protease inhibitor monotherapy as a maintenance strategy: an observational study. AIDS. - 2012. - Vol. 26. - pp. 2345-50.

**Gutmann** C Cusini A, Günthard HF, Fux C, Hirschel B, Decosterd LA, Cavassini M, Yerly S, Vernazza PL. Randomized controlled study demonstrating failure of LPV/r monotherapy in HIV: the role of compartment and CD4-nadir. AIDS. - 2010. - Vol. 24. - pp. 2347-2354...

Jacobson JM Lalezari JP, Thompson MA, Fichtenbaum CJ, Saag MS, Zingman BS, D'Ambrosio P, Stambler N, Rotshteyn Y, Marozsan AJ, Maddon PJ, Morris SA, Olson WC. study of the CCR5 monoclonal antibody PRO 140 administered intravenously to HIV-infected adults. Antimicrob Agents Chemother.. - 2010. - Vol. 54. - pp. 4137-42..

Jacobson JM Saag MS, Thompson MA, Fischl MA, Liporace R, Reichman RC, Redfield RR, Fichtenbaum CJ, Zingman BS, Patel MC, Murga JD, Pemrick SM, D'Ambrosio P, Michael M, Kroger H, Ly H, Rotshteyn Y, Buice R, Morris SA, Stavola JJ, Maddon PJ, Kremer AB, Ols Antiviral activity of single-dose PRO 140, a CCR5 monoclonal antibody, in HIV-infected adults. J Infect Dis.. - 2008. - Vol. 198. - pp. 1345-52..




- **Jacobson JM Thompson MA, Lalezari JP, Saag MS, Zingman BS, D'Ambrosio P, Stambler N, Rotshteyn Y, Marozsan AJ, Maddon PJ, Morris SA, Olson WC.** Anti-HIV-1 activity of weekly or biweekly treatment with subcutaneous PRO 140, a CCR5 monoclonal antibody. J Infect Dis.. 2010. Vol. 201. pp. 1481-7.
- **Katlama** C **Valantin MA**, **Algarte-Genin M**, **et al.** Efficacy of darunavir/ritonavir maintenance monotherapy in patients with HIV-1 viral suppression: a randomized open-label, noninferiority trial MONOI-ANRS 136 AIDS. 2010. Vol. 24. pp. 2365-2374.
- Marozsan A. J., T. Parsons, W. Huang, E. Stawiski, J. M. Whitcomb, P. J. Maddon, and W. C. Olson. Clonal analysis of HIV-1 co-receptor tropism change following treatment with PRO 140, a CCR5 monoclonal antibody. 48th Annual ICAAC / IDSA 46th Annual Meeting. Washington, DC.: [s.n.], 2008. Vols. Abstract H-1218.
- Meynard JL Bouteloup V, Landman R, Bonnard P, Baillat V, Cabie A, Kolta S, Izopet J, Taburet AM, Mercie P, Chene G, Girard PM. Lopinavir/ritonavirmonotherapy versus current treatment continuation for maintenance therapy of HIV-1infection: the KALESOLO trial. J Antimicrob Chemother.. 2010. Vol. 65. pp. 2436-2444.
- Moltó J Santos JR, Negredo E, Miranda C, Videla S, Clotet B. Lopinavir/ritonavir monotherapy as a simplification strategy in routine clinical practice. J Antimicrob Chemother.. 2007. 60. pp. 436-439.
- **Nishikawa M Takashima K, Nishi T, Furuta RA, Kanzaki N, Yamamoto Y et al.** Analysis of binding sites for the new small-molecule CCR5 antagonist TAK-220 on human CCR5. Antimicrob Agents Chemother. 2005. Vol. 49(11). pp. 4708-4715..
- Nunes EP Santini de Oliveira M, Merçon M, Zajdenverg R, Faulhaber JC, Pilotto JH, Ribeiro JE, Norton M, Schechter M. Monotherapy with Lopinavir/Ritonavir as maintenance after HIV-1 viral suppression: results of a 96-week randomized, controlled, open-label, pilot trial (KalMo study). HIV Clin Trials.. 2009. Vol. 10. pp. 368-374..
- Pulido F Arribas JR, Delgado R, Cabrero E, González-García J, Pérez-Elias MJ, Arranz A, Portilla J, Pasquau J, Iribarren JA, Rubio R, Norton M. Lopinavir-ritonavir monotherapy versus lopinavir-ritonavir and two nucleosides for maintenance therapy of HIV. AIDS. 2008. Vol. 22. pp. F1-9.
- Richman D. D., D. Havlir, J. Corbeil, D. Looney, C. Ignacio, S. A. Spector, J. Sullivan, S. Cheeseman, K. Barringer, D. Pauletti. Nevirapine resistance mutations of human immunodeficiency virus type 1 selected during therapy. J Virol.. 1994. Vol. 68. pp. 1660-1666...
- Saag M. S., E. A. Emini, O. L. Laskin, J. Douglas, W. I. Lapidus, W. A. Schleif, R. J. Whitley, C. Hildebrand, V. W. Byrnes, J. C. Kappes. A short-term clinical evaluation of L-697,661, a non-nucleoside inhibitor of HIV-1 reverse transcriptase. N.Engl.J Med.. 1993. Vol. 329. pp. 1065-1072..
- Simioni S Cavassini M, Annoni J, Abraham AR, Bourquin I, Schiffer V, Calmy A, Chave J, Giacobini E, Hirschel B, Du Pasquier RA Cognitive dysfunction in HIV patients despite long-standing suppression of viremia.. 2010. Vol. 24. pp. 1243-1250.




Date: 30-Mar-2021



**Spreen WR Margolis DA, Pottage JC Jr** Long-acting injectable antiretrovirals for HIV treatment and prevention.. - [s.l.]: Curr Opin HIV AIDS., 2013. - Vol. 8(6):565571.

**Thompson M., Lalezari, J., Saag, M., Jacobson, J., Zingman, B., Stambler, N., D'Ambrosio, P., Maddon, P., Olson, W., and Morris, S.** Weekly and bi-weekly subcutaneous PRO 140 demonstrates potent, sustained antiviral activity. 16th Conference on Retroviruses and Opportunistic Infections. - Montreal QE, Canada, : [s.n.], 2009. - Vol. Abstract #571a.

Thompson MA Aberg JA, Hoy JF, Telenti A, Benson C, Cahn P, Eron JJ, Gunthard HF, Hammer SH, Reiss P, Richman DD, Rizzardini G, Thomas DL, Jacobsen DM, Volberding PA. Antiretroviral Treatment of Adult HIV Infection: 2012 Recommendations of the International Antiviral Society—USA Panel JAMA. - 2012. - Vol. 308. - pp. 387-402.


Date: 30-Mar-2021



#### 16 APPENDIX

#### 16.1 APPENDIX I: AIDS-DEFINING CONDITIONS

- Bacterial infections, multiple or recurrent\*
- Candidiasis of bronchi, trachea, or lungs
- Candidiasis of esophagus<sup>†</sup>
- Cervical cancer, invasive§
- Coccidioidomycosis, disseminated or extrapulmonary
- Cryptococcosis, extrapulmonary
- Cryptosporidiosis, chronic intestinal (> 1 month's duration)
- Cytomegalovirus disease (other than liver, spleen, or nodes), onset at age > 1 month
- Cytomegalovirus retinitis (with loss of vision)<sup>†</sup>
- Encephalopathy, HIV related
- Herpes simplex: chronic ulcers (> 1 month's duration) or bronchitis, pneumonitis, or esophagitis (onset at age > 1 month)
- Histoplasmosis, disseminated or extrapulmonary
- Isosporiasis, chronic intestinal (> 1 month's duration)
- Kaposi sarcoma<sup>†</sup>
- Lymphoid interstitial pneumonia or pulmonary lymphoid hyperplasia complex\*†
- Lymphoma, Burkitt (or equivalent term)
- Lymphoma, immunoblastic (or equivalent term)
- Lymphoma, primary, of brain
- *Mycobacterium avium* complex or *Mycobacterium kansasii*, disseminated or extrapulmonary<sup>†</sup>
- *Mycobacterium tuberculosis* of any site, pulmonary, †§ disseminated, † or extrapulmonary †
- *Mycobacterium*, other species or unidentified species, disseminated<sup>†</sup> or extrapulmonary<sup>†</sup>
- Pneumocystis jirovecii pneumonia<sup>†</sup>
- Pneumonia, recurrent<sup>†§</sup>
- Progressive multifocal leukoencephalopathy
- Salmonella septicemia, recurrent
- Toxoplasmosis of brain, onset at age > 1 month<sup>†</sup>




# Wasting syndrome attributed to HIV

Source: http://www.cdc.gov/mmwr/preview/mmwrhtml/rr5710a2.htm


<sup>\*</sup> Only among children aged < 13 years. (CDC. 1994 Revised classification system for human immunodeficiency virus infection in children less than 13 years of age. MMWR 1994;43[No. RR-12].)

<sup>&</sup>lt;sup>†</sup>Condition that might be diagnosed presumptively.

<sup>§</sup> Only among adults and adolescents aged ≥ 13 years. (CDC. 1993 Revised classification system for HIV infection and expanded surveillance case definition for AIDS among adolescents and adults. MMWR 1992;41[No. RR-17].)





# 16.2 APPENDIX II: DIVISION OF AIDS TABLE FOR GRADING THE SEVERITY OF ADULT AND PEDIATRIC ADVERSE EVENTS (DAIDS AE GRADING TABLE)

http://rsc.tech-

 $res.com/Document/safety and pharmacovigilance/DAIDS\_AE\_Grading\_Table\_v2\_NOV2014.pdf$ 




# 16.3 APPENDIX III: ADVERSE EVENTS OF SPECIAL INTEREST: INJECTION SITE REACTIONS

The following table should be used to characterize injection-site reactions and provide appropriate grading of severity (DAIDS and modified additions).

| Injection-site Reactions | | | | |
|---|---|---|---|---|
| Parameter | Grade 1 (Mild) | Grade 2<br>(Moderate) | Grade 3 (Severe) | Grade 4<br>(Potentially life-<br>threatening) |
| Injection-site pain | Pain without<br>touching or pain<br>when area is<br>touched: no or<br>minimal limitation<br>of use of limb | Pain without touching or pain when area is touched limiting use of limb OR causing greater than minimal interference with usual social and functional activities | Pain without<br>touching or pain<br>when area is<br>touched causing<br>inability to perform<br>usual social and<br>functional<br>activities | Pain without touching or pain when area is touched causing inability to perform basic self-care function OR hospitalization (other than emergency room visit) indicated for management of pain/tenderness |
| Characterization of<br>the injection site, if<br>not normal | Erythema OR<br>induration of 5x5<br>cm - 9x9 cm (or 25<br>cm2-81 cm2) | Erythema OR<br>induration OR<br>Edema > 9 cm any<br>diameter (or > 81<br>cm2) | Ulceration OR<br>secondary infection<br>OR Phlebitis or<br>Sterile abscess OR<br>drainage | Necrosis<br>(involving dermis<br>and deeper tissue) |
| Pruritus associated with injection | Itching localized to<br>injection site AND<br>relieved<br>spontaneously or<br>< 48 hours of<br>treatment | Itching beyond the injection site but not generalized OR itching localized to injection site requiring ≥ 48 hours treatment | Generalized itching causing inability to perform usual social and functional activities | N/A |
| Bleeding | Initial bleed that<br>does not exceed<br>bandage and<br>spontaneously<br>stops | Bleeding that<br>exceeds bandage<br>and spontaneously<br>stops | Continued bleeding<br>that requires<br>change of dressing<br>and alternative<br>injection site | N/A |
| Absorption of drug | Minor elevation of<br>skin at injection<br>site but no leakage<br>of injection<br>material | Leakage at injection site ceases with decrease in injection rate | Leakage at injection site that does not cease with decrease in injection rate | |




# 16.4 APPENDIX V: NEUROLOGICAL ASSESSMENT

# Three Question Screening Survey (Simioni, et al, 2010)

- 1. 'Do you experience frequent memory loss (e.g. do you forget the occurrence of special events even the more recent ones, appointments, etc.)'?
- 2. 'Do you feel that you are slower when reasoning, planning activities, or solving problems'?
- 3. 'Do you have difficulties paying attention (e.g. to a conversation, a book, or a movie)'?

For each question, subjects should provide one of the following answers: 'never', 'hardly ever', or 'yes, definitely'.

If subject answers "yes, definitely" to any question, additional neurological assessment modalities may be used as per Investigator's discretion.

